CLINICAL TRIAL: NCT02853435
Title: A Phase I; Multi-Center; Open-Label (Parts 1 and 2); Randomized, Double-Blind, Placebo-Controlled (Part 3); Single-Dose; 3-Part Study to Evaluate the Relative Bioavailability of Three Formulations in Healthy Subjects, Food Effect on Tablet Formulation in Healthy Subjects, and Pharmacokinetics of Gepotidacin (GSK2140944) in Japanese Subjects in Fasted and Fed States
Brief Title: To Assess Bioavailability, Food Effect and Pharmacokinetics of Gepotidacin Tablets: A Phase I, Single-Dose, 2 Part Study in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 117351
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Infections, Bacterial
Keywords: Cross-over; Gepotidacin; Pharmacokinetics; Relative Bioavailability; non-compartmental PK analysis; High shear wet granulation
MeSH Terms: conditions — Bacterial Infections | interventions — gepotidacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part1a: Gepotidacin 1500 mg-Sequence A-capsules, B-RC, C-HSWG (Experimental): Subjects will be receive treatment sequence (ABC) which is a single dose of gepotidacin 1500 mg (three tablets of 500 mg) reference capsule (Treatment A) in Period 1, 1500 mg (two tablets of 750 mg) RC tablet (Treatment B) in Period 2 or 1500 mg (two tablets of 750 mg) HSWG tablet (Treatment C) in Period 3, according to randomization. There will be a washout period of at least 3 days between doses.
  Interventions: Drug: Gepotidacin RC Tablet; Drug: Gepotidacin HSWG Tablet; Drug: Gepotidacin Capsule
- Part1a: Gepotidacin 1500 mg-Sequence C-HSWG, A-capsules, B-RC) (Experimental): Subjects will receive treatment sequence (CAB) to receive a single dose of gepotidacin 1500 mg (two tablets of 750 mg) HSWG tablet (Treatment C) in Period 1, 1500 mg (three tablets of 500 mg) reference capsule (Treatment A) in Period 2 or 1500 mg (two tablets of 750 mg) RC tablet (Treatment B) in Period 3 according to randomization. There will be a washout period of at least 3 days between doses.
  Interventions: Drug: Gepotidacin RC Tablet; Drug: Gepotidacin HSWG Tablet; Drug: Gepotidacin Capsule
- Part1a: Gepotidacin 1500 mg-Sequence B-RC, C-HSWG, A-capsules) (Experimental): Subjects will receive treatment sequence (BCA) to receive a single dose of gepotidacin 1500 mg (two tablets of 750 mg) RC tablet (Treatment B) in period 1, 1500 mg (two tablets of 750 mg) HSWG tablet (Treatment C) in Period 2, or 1500 mg (three tablets of 500 mg) (Treatment A) in Period 3 reference capsule according to randomization.. There will be a washout period of at least 3 days between doses.
  Interventions: Drug: Gepotidacin RC Tablet; Drug: Gepotidacin HSWG Tablet; Drug: Gepotidacin Capsule
- Part1b: Gepotidacin 1500 mg-Sequence DE-fasted followed by fed (Experimental): Subjects will receive treatment sequence (DE) according to randomization which is a single 1500 mg (two tablets of 750 mg) dose of gepotidacin tablet (RC or HSWG) selected from Part 1a under fasted condition (Treatment D) in Period 1 followed by fed conditions (Treatment E) in period 2. There will be a washout period of at least 3 days between doses.
  Interventions: Drug: Gepotidacin RC Tablet; Drug: Gepotidacin HSWG Tablet
- Part1b: Gepotidacin 1500 mg-Sequence ED-fed followed by fasted (Experimental): Subjects will be receive treatment sequence (ED) according to randomization which is single 1500 mg (two tablets of 750 mg) dose of gepotidacin tablet (RC or HSWG) selected from Part 1a under fed condition (Treatment E) in period 1 followed by fasted conditions (Treatment D) in Period 2. There will be a washout period of at least 3 days between doses.
  Interventions: Drug: Gepotidacin RC Tablet; Drug: Gepotidacin HSWG Tablet
- Part 2a: Gepotidacin 1500 mg (RC or HSWG)- Japanese subjects (Experimental): Japanese subjects will receive a single 1500 mg (two tablets of 750 mg) dose of gepotidacin tablet (RC or HSWG) selected from Part 1a.
  Interventions: Drug: Gepotidacin RC Tablet; Drug: Gepotidacin HSWG Tablet
- Part 2b: Gepotidacin 1500 mg (RC or HSWG)- Chinese subjects (Experimental): Chinese subjects will receive a single 1500 mg (two tablets of 750 mg) dose of gepotidacin tablet (RC or HSWG) selected from Part 1a.
  Interventions: Drug: Gepotidacin RC Tablet; Drug: Gepotidacin HSWG Tablet

INTERVENTIONS:
Drug: Gepotidacin RC Tablet — The tablet is a capsule shape white film coated tablet with no identifying markings. This is an immediate release tablet containing gepotidacin 750 mg (free base) and inactive formulation excipients administered orally with 240 mL of water. Up to an additional 100 mL of water may be given to assist in swallowing tablets.
Drug: Gepotidacin HSWG Tablet — The tablet is an oval shape white film coated tablet with no identifying markings. This is an immediate release tablets containing gepotidacin 750 mg (free base) and inactive formulation excipients administered orally with 240 mL of water. Up to an additional 100 mL of water may be given to assist in swallowing tablets.
Drug: Gepotidacin Capsule — It is a pink gelatin size 00 capsule with no identifying markings containing slightly agglomerated pale yellow to grayish yellow to yellowish gray powder. This is an immediate release capsules containing gepotidacin 500 mg (mesylate salt) and inactive formulation excipients administered orally with 240 mL of water. Up to an additional 100 mL of water may be given to assist in swallowing capsules.
  Arms: Part1a: Gepotidacin 1500 mg-Sequence A-capsules, B-RC, C-HSWG; Part1a: Gepotidacin 1500 mg-Sequence B-RC, C-HSWG, A-capsules); Part1a: Gepotidacin 1500 mg-Sequence C-HSWG, A-capsules, B-RC)

SUMMARY:
This study is divided in 2 parts. Part 1a is being conducted to evaluate the safety, tolerability, and relative bioavailability of the 2 free base tablet formulations (roller compacted [RC] and high shear wet granulation [HSWG]) compared to the reference capsule formulation under fasted conditions. This is a 3-period; cross-over study that will guide which gepotidacin formulation will be used for future studies. Following review of pharmacokinetic (PK) and safety data in Part 1a, a decision will be made whether to proceed with Parts 1b and 2.

Part 1b is a 2-period, cross-over study and will assess the effect of food on the PK of the selected gepotidacin tablet formulation from Part 1a. In Part 2, the PK of the selected gepotidacin tablet formulation from Part 1a in Japanese (2a) and Chinese (2b) subjects will be evaluated under fasted conditions.

The duration of the study (from Screening to the Follow-up visit) will be approximately 44 days (Part 1a), 41 days (Part 1b) and 38 days (Part 2a and 2b each), respectively. The approximate number of subjects enrolled in Part 1a will be 27 (9 subjects in each of the 3 treatment sequences), 16 in Part 1b (8 subjects in each of the 2 treatment sequences) and 12 Japanese and 12 Chinese subjects in Part 2a and 2b, respectively.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects between 18 and 64 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator based on medical history, clinical laboratory results (serum chemistry, hematology, urinalysis, and serology), vital sign measurements, 12-lead ECG results, and physical examination findings. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Additional inclusion criteria for Japanese subjects (Part 2a only): the subject was a non-naturalized Japanese citizen and held a Japanese passport, the subject had 2 Japanese parents and 4 Japanese grandparents who were all non naturalized Japanese citizens, as confirmed by interview and the subject had been living outside of Japan for up to 10 years as confirmed by interview.
* Additional inclusion criteria for Chinese subjects (Part 2b only): the subject was a non-naturalized Chinese citizen and held a Chinese passport, the subject had 2 Chinese parents and 4 Chinese grandparents who were all non naturalized Chinese citizens, as confirmed by interview, the subject had been living outside of China for up to 10 years as confirmed by interview.
* Body weight for subjects in Part 1a and 1b: more than equal to (>=) 50 kilogram (kg) and body mass index (BMI) within the range 19 and 32 kilogram per meter square (kg/m^2), inclusive and for Japanese and Chinese subjects (Part 2a and 2b): >=50 kg and BMI within the range 18 and 32 kg/m^2, inclusive.
* Male or female: a female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin test, not lactating, and at least one of the following conditions applies. Non-reproductive potential defined as: pre-menopausal females with one of the following: documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, documented bilateral oophorectomy and postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle-stimulating hormone and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential from 30 days prior to the first dose of study medication and until completion of the Follow-up visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria

* Subject has a clinically significant abnormality in past medical history or at the Screening physical examination that in the investigator's opinion may place the subject at risk or interfere with outcome variables of the study. This includes, but is not limited to, history or current cardiac, hepatic, renal, neurologic, gastrointestinal, respiratory, hematologic, or immunologic disease.
* Subject has any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug, or any other condition that may place the subject at risk, in the opinion of the investigator.
* QTc more than (>) 450 millisecond (msec).
* Use of a systemic antibiotic within 30 days of Screening.
* Within 2 months before Screening, either a confirmed history of Clostridium difficile diarrhea infection or a past positive Clostridium difficile toxin test.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinic uses heparin to maintain intravenous cannula patency).
* Subjects cannot use any over-the-counter, or prescription medication (except for hormonal contraceptives and/or acetaminophen), vitamin supplement, or herbal medication within 7 days (or 5 half-lives, whichever is longer) before dosing and during the study.
* History of regular alcohol consumption within 6 months of screening defined as an average weekly intake of >21 units (or an average daily intake of >3 units) for males or an average weekly intake of >14 units (or an average daily intake >2 units) for females. One unit is equivalent to 270 milliliter (mL) of full strength beer, 470 mL of light beer, 30 mL of spirits, or 100 mL of wine.
* Urinary cotinine level indicative of smoking or history or regular use of tobacco- or nicotine containing products within 3 months before screening.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen, positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Female subject has a positive pregnancy test result or is lactating at Screening or upon admission to the clinic.
* ALT >1.5×upper limit of normal (ULN)
* Bilirubin >1.5×ULN (isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin less than [<] 35 percent [%]).
* Urinalysis positive for blood without other cause identified.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus antibody.
* Subject has clinically significant abnormal findings in serum chemistry, hematology, or urinalysis results obtained at Screening or Day -1.
* Donation of blood in excess of 500 mL within 12 weeks prior to dosing or participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Previous exposure to gepotidacin within 12 months prior to the first dosing day.
* Exclusion criteria for screening and baseline 12-lead ECG (a single repeat is allowed for eligibility determination): male subjects with heart rate <40 and >100 beats per minute (bpm), female subjects with heart rate <50 and >100 bpm, PR interval <120 and >220 msec for male and female subjects, QRS duration <70 and >120 msec in both male and female subjects and corrected QT interval using Bazett's formula (QTcB) or corrected QT interval using Fridericia's formula (QTcF) >450 msec in both male and female subjects. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block [second degree or higher], Wolf Parkinson White syndrome), sinus pauses >3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GlaxoSmithKline medical monitor, will interfere with the safety of the individual subject.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Subject is unable to comply with all study procedures, in the opinion of the investigator.
* The subject should not participate in the study, in the opinion of the investigator or sponsor.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Austin, Texas

REFERENCES:
- [Derived] Barth A, Hossain M, Brimhall DB, Perry CR, Tiffany CA, Xu S, Dumont EF. Pharmacokinetics of Oral Formulations of Gepotidacin (GSK2140944), a Triazaacenaphthylene Bacterial Type II Topoisomerase Inhibitor, in Healthy Adult and Adolescent Participants. Antimicrob Agents Chemother. 2022 Jan 18;66(1):e0126321. doi: 10.1128/AAC.01263-21. Epub 2021 Oct 11. PMID 34633853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 2 centers in the United States from 04-August-2016 to 18-October-2017. Since the relative bio-availability of the roller compacted(RC) tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Pre-assignment Details: A total of 48 participants were enrolled in the study of which 26 participants were randomized in Part 1a, 10 participants were randomized in Part 2 and 12 participants were part of Placebo-controlled Part 3.
Groups:
- Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG: Participants received gepotidacin 1500 milligrams (mg) (3 x 500 mg) (Reference [R]) capsules in treatment period 1 followed by gepotidacin 1500 mg (2 x 750 mg) related RC tablets in treatment period 2 followed by gepotidacin 1500 mg (2 x 750 mg) high shear wet granulation (HSWG) tablets orally for 3 days in each treatment period in Part 1a. There was a washout period of at least 3 days between the doses.
- Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC: Participants received gepotidacin 1500 mg (2 x 750 mg) HSWG tablets in treatment period 1 followed by gepotidacin 1500 mg (3 x 500 mg) - R capsules in treatment Period 2 followed by gepotidacin 1500 mg (2 x 750 mg) RC tablets in treatment period 3 orally for 3 days in each treatment period in Part 1a. There was a washout period of at least 3 days between the doses.
- Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R: Participants received gepotidacin 1500 mg (2 x 750 mg) RC tablets in treatment period 1 followed by gepotidacin 1500 mg (2 x 750 mg) HSWG tablets in treatment period 2 followed by gepotidacin 1500 mg (3 x 500 mg) - R capsules in treatment period 3 for 3 days in each treatment period in Part 1a. There was a washout period of at least 3 days between the doses.
- Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC: Participants received gepotidacin 1500 mg (2 x 750 mg) RC tablets in treatment period 1 followed by gepotidacin 3000 mg (4 x 750 mg) RC tablets in treatment period 2 orally for 3 days in each treatment period in Part 2. There was a washout period of at least 3 days between the doses.
- Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000: Participants received gepotidacin 1500 mg (2 x 750 mg) RC tablets - fed in treatment period 1 followed by Gepotidacin 2250 mg (3 x 750 mg) RC tablets - fed in treatment period 2 followed by Gepotidacin 2250 mg (3 x 750 mg) RC tablets - fed in treatment period 3 orally for 3 days in each treatment period in part 3. There was a washout period of at least 3 days between the doses.
- Placebo Then Placebo Then Placebo: Participants received matching placebo to gepotidacin 1500 mg RC tablets in treatment period 1 followed by matching placebo to gepotidacin 2250 mg in treatment period 2 followed by matching placebo to gepotidacin 2250 mg RC tablets in treatment period 3 orally for 3 days in each treatment Period in Part 3. There was a washout period of at least 3 days between the doses.
Period: Part 1a, Period 1 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 9 | 9 | 8 | 0 | 0 | 0
Completed | 9 | 9 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1a, Washout Period 1 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 9 | 9 | 8 | 0 | 0 | 0
Completed | 9 | 9 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1a, Period 2 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 9 | 9 | 8 | 0 | 0 | 0
Completed | 9 | 9 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1a, Washout Period 2 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 9 | 9 | 8 | 0 | 0 | 0
Completed | 9 | 9 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1a, Period 3 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 9 | 9 | 8 | 0 | 0 | 0
Completed | 9 | 9 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 1 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 10 | 0 | 0
Completed | 0 | 0 | 0 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 1 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 10 | 0 | 0
Completed | 0 | 0 | 0 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 2 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 10 | 0 | 0
Completed | 0 | 0 | 0 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Period 1 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 0 | 10 | 2
Completed | 0 | 0 | 0 | 0 | 10 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Washout Period 1 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 0 | 10 | 2
Completed | 0 | 0 | 0 | 0 | 10 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Period 2 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 0 | 10 | 2
Completed | 0 | 0 | 0 | 0 | 10 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Washout Period 2 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 0 | 10 | 2
Completed | 0 | 0 | 0 | 0 | 9 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 3, Period 3 (3 Days)
Arm/Group | Gepotidacin-R Then Gepotidacin RC Then Gepotidacin HSWG | Gepotidacin HSWG Then Gepotidacin- R Then Gepotidacin RC | Gepotidacin-RC Then Gepotidacin HSWG Then Gepotidacin-R | Gepotidacin 1500 mg RC Then Gepotidacin 3000 mg RC | Gepotidacin 1500 Then Gepotidacin 2250 Then Gepotidacin 3000 | Placebo Then Placebo Then Placebo
Started | 0 | 0 | 0 | 0 | 9 | 2
Completed | 0 | 0 | 0 | 0 | 9 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Participants-Part 1a: Participants received gepotidacin 1500 mg (3 x 500 mg) capsules, gepotidacin 1500 mg (2 x 750 mg) RC tablets and gepotidacin 1500 mg (2 x 750 mg) HSWG tablets orally in one of the 3 treatment periods in a cross-over manner. There was a washout period of at least 3 days between the doses.
- Total Participants-Part 2: Participants received gepotidacin 1500 mg (2 x 750 mg) RC tablets and gepotidacin 3000 mg (4 x 750 mg) RC tablets orally in one of the 2 treatment periods in a cross-over manner. There was a washout period of at least 3 days between the doses.
- Total Participants- Part 3: Participants received gepotidacin 1500 mg (2 x 750 mg) RC tablets - fed, gepotidacin 2250 mg (3 x 750 mg) RC tablets - fed and gepotidacin 3000 mg (4 x 750 mg) RC tablets - fed orally in one of the 3 treatment periods in a cross-over manner. There was a washout period of at least 3 days between the doses.
- Total: Total of all reporting groups
Arm/Group | Total Participants-Part 1a | Total Participants-Part 2 | Total Participants- Part 3 | Total
Number analyzed (Participants) | 26 | 10 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (10.64) | 55.6 (6.43) | 37.8 (7.93) | 42.5 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 6 | 19
  Male | 21 | 2 | 6 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 10 | 0 | 0 | 10
  White - White/Caucasian/European Heritage | 16 | 0 | 0 | 16
  Asian - Japanese Heritage | 0 | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 (Pre-dose) Extrapolated to Infinite Time (AUC [0-infinity]) of Plasma Gepotidacin for Part 1a
Description: Blood samples for pharmacokinetic (PK) analysis of gepotidacin were collected at Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 1a. For each sample, 3 milliliters (mL) of blood was drawn via an indwelling catheter and/or direct venipuncture into tubes containing ethylenediaminetetraacetate anticoagulant. PK parameters were determined from the plasma concentration-time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher. The PK Parameter Population consisted of all participants in the PK Population, for whom valid and evaluable PK parameters were derived. Statistics has been presented on geometric least square (LS) means.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in each treatment period
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Groups:
- Gepotidacin 1500 mg - R Capsules: Participants received gepotidacin 1500 (3 x 500) mg - R capsules orally in one of the 3 treatment periods for 3 days in Part 1a.
- Gepotidacin 1500 mg RC Tablets: Participants received gepotidacin 1500 (2 x 750) mg RC tablets orally in one of the 3 treatment periods for 3 days in Part 1a.
- Gepotidacin 1500 mg HSWG Tablets: Participants received gepotidacin 1500 mg (2 x 750 mg) HSWG tablets orally in one of the 3 treatment periods in Part 1a.
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
hours*nanograms/milliliter | 16733 (25.7) | 17495 (23.0) | 18646 (24.0)
Statistical Analysis 1: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg RC Tablets; Test type: Other; Ratio of geometric LS means = 1.0417, 90% CI 2-sided [0.9809 to 1.1063] — A mixed effects model with treatment, sequence, period as fixed effects and participant within sequence as random effect was performed on the natural log-transformed parameters AUC(0-inf)
Statistical Analysis 2: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg HSWG Tablets; Test type: Other; Ratio of geometric LS means = 1.1108, 90% CI 2-sided [1.0459 to 1.1797] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time 0 (Pre-dose) to Time of the Last Quantifiable Concentration (AUC [0-t]) of Plasma Gepotidacin for Part 1a
Description: Blood samples for PK analysis of gepotidacin were collected at Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 1a. For each sample, 3 mL of blood was drawn via an indwelling catheter and/or direct venipuncture into tubes containing ethylenediaminetetraacetate anticoagulant. PK parameters were determined from the plasma concentration-time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
hours*nanograms/milliliters | 16409 (26.2) | 17125 (23.4) | 18317 (24.1)
Statistical Analysis 1: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg RC Tablets; Test type: Other; Ratio of geometric LS means = 1.0408, 90% CI 2-sided [0.9792 to 1.1062] — A mixed effects model with treatment, sequence, period as fixed effects and participant within sequence as random effect was performed on the natural log-transformed parameters AUC(0-t)
Statistical Analysis 2: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg HSWG Tablets; Test type: Other; Ratio of geometric LS means = 1.1138, 90% CI 2-sided [1.0479 to 1.1838] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Relative Bioavailability of Drug (Frel) of Plasma Gepotidacin for Part 1a
Description: Blood samples for PK analysis of gepotidacin were collected at Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 1a. For each sample, 3 mL of blood was drawn via an indwelling catheter and/or direct venipuncture into tubes containing ethylenediaminetetraacetate anticoagulant. PK parameters were determined from the plasma concentration-time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher. NA indicates data was not available as this was the reference capsule the Frel of each tablet type was being compared to.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC (0-infinity)
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
Ratio of AUC (0-infinity) | NA (NA) — This was the reference capsule the Frel of each tablet was being compared to. | 1.05 (22.3) | 1.11 (16.5)

4. Primary Outcome: Maximum Observed Concentration (Cmax) Determined Directly From the Concentration Time Data of Plasma Gepotidacin for Part 1a
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
nanograms/milliliter | 4648 (43.8) | 4487 (43.6) | 5349 (46.8)
Statistical Analysis 1: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg RC Tablets; Test type: Other; Ratio of geometric LS means = 0.9586, 90% CI 2-sided [0.8440 to 1.0888] — A mixed effects model with treatment, sequence, period as fixed effects and participant within sequence as random effect was performed on the natural log-transformed parameters Cmax
Statistical Analysis 2: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg HSWG Tablets; Test type: Other; Ratio of geometric LS means = 1.1487, 90% CI 2-sided [1.0113 to 1.3047] — [estimate comment as in outcome 4, analysis 1]

5. Primary Outcome: Time to First Occurrence of Cmax (Tmax) of Plasma Gepotidacin for Part 1a
Description: Blood samples for PK analysis of gepotidacin were collected at Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 1a. For each sample, 3 mL of blood was drawn via an indwelling catheter and/or direct venipuncture into tubes containing ethylenediaminetetraacetate anticoagulant. PK parameters were determined from the plasma concentration-time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
hours | 1.50 [1.00 to 4.00] | 1.50 [0.50 to 4.00] | 1.00 [0.50 to 3.00]
Statistical Analysis 1: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg RC Tablets; Test type: Other; p = 0.309, Wilcoxon signed-rank test. — The p-value is from Wilcoxon signed-rank test; Median Difference (Final Values) = -0.233, 90% CI 2-sided [-0.267 to 0.000] — The median, median difference and 90% CI of the median difference are from Hodge-Lehmann estimate
Statistical Analysis 2: Comparison: Gepotidacin 1500 mg - R Capsules vs Gepotidacin 1500 mg HSWG Tablets; Test type: Other; p < 0.001, Wilcoxon signed-rank test. — The p-value is from Wilcoxon signed-rank test; Median Difference (Final Values) = -0.492, 90% CI 2-sided [-0.500 to -0.250] — The median, median difference and 90% CI of the median difference are from Hodge-Lehmann estimate

6. Primary Outcome: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) of Plasma Gepotidacin for Part 1a
Description: as for outcome 5
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
hours | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.50]

7. Primary Outcome: Terminal Phase Half-life (t1/2) of Plasma Gepotidacin for Part 1a
Description: as for outcome 5
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
hours | 10.29 (13.7) | 10.24 (15.2) | 10.24 (12.1)

8. Primary Outcome: Total Unchanged Drug (Total Amount of Drug Excreted in Urine [Ae Total]) for Part 1a
Description: PK urine samples were collected at 0 (predose), 0 to 2, 2 ot 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48 hours. PK parameters were determined from the urine concentration- time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
milligrams | 274.925 (28.6) | 286.751 (22.2) | 284.510 (30.0)

9. Primary Outcome: Percentage of the Given Dose of Drug Excreted in Urine (fe%) of Plasma Gepotidacin for Part 1a
Description: PK urine samples were collected at 0 (pre-dose), 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48 hours. PK parameters were determined from the urine concentration- time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage dose of drug excreted
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
Percentage dose of drug excreted | 18.329 (28.6) | 19.116 (22.2) | 18.968 (30.0)

10. Primary Outcome: Renal Clearance of Drug in Urine (CLr) for Part 1a
Description: as for outcome 9
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
liters/hour | 16.761 (21.7) | 16.740 (19.6) | 15.532 (22.3)

11. Primary Outcome: Amount of Drug Excreted in Urine in a Time Intervals for Pre-dose, 0 to 2 Hours, 2 to 4 Hours, 4 to 6 Hours, 6 to 8 Hours, 8 to 12 Hours, 12 to 24 Hours, 24 to 36 Hours, and 36 to 48 Hours (Ae [t1-t2]) for Part 1a
Description: PK urine samples were collected at 0 (pre-dose), 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48 hours. PK parameters were determined from the urine concentration- time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher. Only those participants available at the specific time points were analyzed (represented by n = X in the category titles).
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
milligrams
  Ae (0-2), n=26,25,26: number analyzed (Participants) | 26 | 25 | 26
  Ae (0-2), n=26,25,26 | 65.817 (95.1) | 60.915 (102.9) | 85.584 (67.7)
  Ae (2-4),n=26,24,25: number analyzed (Participants) | 26 | 24 | 25
  Ae (2-4),n=26,24,25 | 72.734 (67.3) | 77.650 (33.6) | 67.419 (72.0)
  Ae (4-6),n=25,25,26: number analyzed (Participants) | 25 | 25 | 26
  Ae (4-6),n=25,25,26 | 36.019 (44.2) | 45.313 (61.1) | 39.361 (39.1)
  Ae (6-8),n=25,26,26: number analyzed (Participants) | 25 | 26 | 26
  Ae (6-8),n=25,26,26 | 22.817 (37.4) | 26.061 (24.9) | 22.755 (28.7)
  Ae (8-12),n=26,26,26 | 21.515 (57.3) | 25.609 (27.7) | 16.590 (75.5)
  Ae (12-24),n=26,26,26 | 19.224 (60.4) | 22.536 (26.9) | 19.432 (32.9)
  Ae (24-36),n=26,26,26 | 8.145 (35.0) | 9.787 (27.8) | 8.185 (44.4)
  Ae (36-48),n=26,26,26 | 4.633 (31.4) | 4.517 (57.7) | 4.319 (41.0)

12. Primary Outcome: Area Under the Urine Concentration-time Curve Over Time 0 (Pre-dose) to 12 Hours (AUC [0-12]) for Part 1a
Description: as for outcome 9
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
micrograms*hours/milliliter | 1904 (82.7) | 1948 (61.2) | 2156 (74.8)

13. Primary Outcome: Area Under the Urine Concentration-time Curve Over Time 0 (Pre-dose) to 24 Hours (AUC [0-24]) After Dosing for Part 1a
Description: as for outcome 9
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 262
micrograms*hours/milliliter | 2373 (74.9) | 2464 (56.3) | 2599 (69.0)

14. Primary Outcome: Area Under the Urine Concentration-time Curve Over Time 0 (Pre-dose) to 48 Hours (AUC [0-48]) After Dosing for Part 1a
Description: PK urine samples were collected at 0 (pre-dose), 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48 hours. PK parameters were determined from the urine concentration- time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher. Only those participants with data available at the indicated time point were analyzed.
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 23 | 26 | 24
micrograms*hours/milliliter | 2597 (69.5) | 2725 (54.4) | 2768 (64.0)

15. Primary Outcome: AUC (0-infinity) of Plasma Gepotidacin for Part 1b
Description: Blood samples for PK analysis of gepotidacin was planned to be collected at Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 1b. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: as for outcome 1
Population: PK Parameter Population. The relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Groups:
- Gepotidacin 1500 mg RC Tablets-fasted: Participants received Gepotidacin 1500 mg (2 x 750 mg) RC tablets orally in the fasted state in one of the 2 treatment periods for 3 days in Part 1b.
- Gepotidacin 3000 mg RC Tablets-fed: Participants received Gepotidacin 1500 mg (2 x 750 mg) RC tablets orally in the fed state in one of the 2 treatment periods for 3 days in Part 1b.
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: AUC (0-t) of Plasma Gepotidacin for Part 1b
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 15
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Cmax of Plasma Gepotidacin for Part 1b
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 15
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Tmax of Plasma Gepotidacin for Part 1b
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 15
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Tlag of Plasma Gepotidacin for Part 1b
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 15
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: t1/2 of Plasma Gepotidacin for Part 1b
Description: as for outcome 15
Time Frame: as for outcome 1
Population: as for outcome 15
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: AUC (0-infinity) of Plasma Gepotidacin for Part 2
Description: Blood samples for PK analysis of gepotidacin were collected at Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 2. For each sample, 3 mL of blood was drawn via an indwelling catheter and/or direct venipuncture into tubes containing ethylenediaminetetraacetate anticoagulant. PK parameters were determined from the plasma concentration-time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Groups:
- Gepotidacin RC 1500 mg Tablets: Participants received a single dose gepotidacin 1500 mg (2 x 750 mg) RC tablets orally in Part 2 Period 1.
- Gepotidacin RC 3000 mg Tablets: Participants received a single dose gepotidacin 3000 mg (4 x 750 mg) RC tablets orally in Part 2 Period 2.
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
hours*nanograms/milliliter | 23137 (34.1) | 46537 (20.9)

22. Primary Outcome: AUC (0-t) of Plasma Gepotidacin for Part 2
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
hours*nanograms/milliliter | 22777 (34.4) | 46120 (21.1)

23. Primary Outcome: Cmax of Plasma Gepotidacin for Part 2
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
nanograms/milliliter | 9177 (94.8) | 15335 (28.6)

24. Primary Outcome: Tlag of Plasma Gepotidacin for Part 2
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
hours | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

25. Primary Outcome: Tmax of Plasma Gepotidacin for Part 2
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
hours | 1.00 [0.50 to 2.00] | 0.56 [0.50 to 2.50]

26. Primary Outcome: t1/2 of Plasma Gepotidacin for Part 2
Description: as for outcome 21
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
hours | 10.73 (10.9) | 8.81 (8.4)

27. Primary Outcome: Total Unchanged Drug (Ae Total) for Part 2
Description: as for outcome 9
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
milligrams | 203.853 (38.8) | 546.263 (51.8)

28. Primary Outcome: Ae (t1-t2) for Part 2
Description: as for outcome 9
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Groups:
- Gepotidacin RC 1500 mg Tablets: Participants received a single dose gepotidacin 1500mg (2 x 750 mg) RC tablets orally in Part 2 Period 1.
- Gepotidacin RC 3000 mg Tablets: Participants received a single dose gepotidacin 3000mg (4 x 750 mg) RC tablets orally in Part 2 Period 2
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
milligrams
  Ae (0-2) | 50.893 (289.7) | 115.793 (73.0)
  Ae (2-4) | 47.995 (42.7) | 131.013 (92.1)
  Ae (4-6) | 21.381 (47.5) | 97.651 (139.4)
  Ae (6-8) | 11.759 (88.2) | 40.670 (36.2)
  Ae (8-12) | 12.519 (104.6) | 29.474 (96.0)
  Ae (12-24) | 9.810 (226.4) | 30.849 (83.9)
  Ae (24-36) | 3.710 (111.0) | 9.754 (51.0)
  Ae (36-48) | 2.743 (114.7) | 3.652 (136.1)

29. Primary Outcome: AUC (0-12) for Part 2
Description: as for outcome 9
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
micrograms*hours/milliliter | 1298 (110.8) | 4758 (64.6)

30. Primary Outcome: AUC (0-24) for Part 2
Description: as for outcome 9
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
micrograms*hours/milliliter | 1714 (88.8) | 5594 (61.9)

31. Primary Outcome: AUC (0-48) for Part 2
Description: PK urine samples were collected at pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48 hours. PK parameters were determined from the urine concentration- time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
micrograms*hours/milliliter | 1875 (83.6) | 5845 (61.1)

32. Primary Outcome: fe% for Part 2
Description: as for outcome 31
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage dose of drug excreted
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
Percentage dose of drug excreted | 13.591 (38.8) | 18.207 (51.8)

33. Primary Outcome: CLr for Part 2
Description: PK urine samples were collected at pre-dose), 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48 hours. PK parameters were determined from the urine concentration- time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
liters/hour | 8.950 (41.5) | 11.834 (32.0)

34. Primary Outcome: AUC (0-infinity) of Plasma Gepotidacin for Part 3
Description: Blood samples for PK analysis of gepotidacin were collected at Pre-dose, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 3. For each sample, 3 mL of blood was drawn via an indwelling catheter and/or direct venipuncture into tubes containing ethylenediaminetetraacetate anticoagulant. PK parameters were determined from the plasma concentration-time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Groups:
- Gepotidacin RC 1500 mg Fed: Participants received a single dose gepotidacin 1500 mg (2 x 750 mg) RC tablets in the fed state orally in Part 3 Period 1.
- Gepotidacin RC 2250 mg Fed: Participants received a single dose gepotidacin 2250 mg (3 x 750 mg) RC tablets in the fed state orally in Part 3 Period 2.
- Gepotidacin RC 3000 mg Fed: Participants received a single dose gepotidacin 3000 mg (4 x 750 mg) RC tablets in the fed state orally in Part 3 Period 3.
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
hours*nanograms/milliliter | 22921 (19.9) | 37235 (17.2) | 50178 (21.9)

35. Primary Outcome: AUC (0-t) of Plasma Gepotidacin for Part 3
Description: Blood samples for PK analysis of gepotidacin were collected at Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours (Day 1), 24, 36 hours (Day 2) and 48 hours (Day 3) in Part 3. For each sample, 3 mL of blood was drawn via an indwelling catheter and/or direct venipuncture into tubes containing ethylenediaminetetraacetate anticoagulant. PK parameters were determined from the plasma concentration-time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher.
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
hours*nanograms/milliliter | 22709 (20.0) | 36938 (17.2) | 49789 (21.7)

36. Primary Outcome: Cmax of Plasma Gepotidacin for Part 3
Description: as for outcome 35
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
nanograms/milliliter | 6502 (27.7) | 9812 (21.1) | 12889 (21.1)

37. Primary Outcome: Tmax of Plasma Gepotidacin for Part 3
Description: as for outcome 35
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
hours | 2.25 [1.00 to 4.00] | 2.05 [1.50 to 4.00] | 2.00 [1.00 to 3.00]

38. Primary Outcome: Tlag of Plasma Gepotidacin for Part 3
Description: as for outcome 35
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
hours | 0.50 [0.00 to 0.50] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

39. Primary Outcome: t1/2 of Plasma Gepotidacin for Part 3
Description: as for outcome 35
Time Frame: as for outcome 1
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
hours | 9.23 (9.7) | 8.19 (7.2) | 7.93 (10.6)

40. Primary Outcome: Total Unchanged Drug (Ae Total) for Part 3
Description: as for outcome 31
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
milligrams | 390.099 (34.3) | 613.635 (32.2) | 895.556 (27.8)

41. Primary Outcome: Urine Ae (t1-t2) for Part 3
Description: PK urine samples were collected at pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48 hours. PK parameters were determined from the urine concentration- time data and were calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.2.1 or higher. Only those participants available at the specific time points were analyzed (represented by n = X in the category titles).
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
milligrams
  Ae (0-2), n=10,10,9 | 27.763 (536.8) | 54.827 (264.1) | 142.546 (96.7)
  Ae (2-4), n=10,10,9 | 132.423 (67.6) | 247.448 (45.5) | 333.805 (43.0)
  Ae (4-6),n=9,10,9: number analyzed (Participants) | 9 | 10 | 9
  Ae (4-6),n=9,10,9 | 63.314 (61.4) | 113.386 (36.9) | 175.739 (36.5)
  Ae (6-8),n=10,10,9 | 54.631 (57.4) | 48.536 (93.3) | 70.582 (70.7)
  Ae (8-12),n=10,10,9 | 35.322 (37.1) | 48.906 (41.0) | 47.392 (85.2)
  Ae (12-24),n=10,10,9 | 14.201 (40.3) | 22.931 (65.9) | 36.214 (65.8)
  Ae (24-36),n=10,10,9 | 6.510 (49.0) | 8.463 (55.4) | 12.642 (50.7)
  Ae (36-48),n=10,10,8: number analyzed (Participants) | 10 | 10 | 8
  Ae (36-48),n=10,10,8 | 3.265 (53.3) | 3.150 (71.5) | 5.641 (42.4)

42. Primary Outcome: Urine AUC (0-12) for Part 3
Description: as for outcome 31
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
micrograms*hours/milliliter | 1573 (48.3) | 2812 (42.4) | 3517 (52.4)

43. Primary Outcome: Urine AUC (0-24) for Part 3
Description: as for outcome 31
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
micrograms*hours/milliliter | 1879 (51.8) | 3301 (45.5) | 4197 (54.1)

44. Primary Outcome: Urine AUC (0-48) for Part 3
Description: as for outcome 31
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
micrograms*hours/milliliter | 2024 (54.3) | 3455 (46.6) | 4390 (54.1)

45. Primary Outcome: fe% for Part 3
Description: as for outcome 31
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage dose of drug excreted
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
Percentage dose of drug excreted | 26.008 (34.3) | 27.273 (32.2) | 29.858 (27.8)

46. Primary Outcome: CLr for Part 3
Description: as for outcome 31
Time Frame: Pre-dose, 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, and 36 to 48 hours.
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed
Number analyzed (Participants) | 10 | 10 | 9
liters/hour | 17.196 (24.8) | 16.598 (26.5) | 17.969 (21.2)

47. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs) for Part 1a
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Participants with non-serious AEs and SAEs has been reported. Safety Population comprised of all participants who received at least 1 dose of study medication and had at least 1 post dose safety assessment.
Time Frame: Up to 14 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Gepotidacin 1500 mg HSWG Tablets: Participants received gepotidacin 1500 mg (2 x 750 mg) HSWG tablets orally in one of the three treatment periods in Part 1a.
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
Participants
  Non serious AE | 8 | 5 | 9
  SAE | 0 | 0 | 0

48. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Glucose, Serum Calcium, Serum Carbon Dioxide, Serum Chloride, Serum Potassium, Serum Sodium and Serum Urea Nitrogen for Part 1a
Description: Blood samples were collected for the assessment of chemistry parameters namely serum glucose, serum calcium, serum carbon dioxide, serum chloride, serum potassium, serum sodium and serum urea nitrogen for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
millimoles/liter
  Serum glucose, Day 3 (48 hour), n=26, 26, 26 | 0.010 (0.2837) | 0.049 (0.3253) | 0.094 (0.2699)
  Serum glucose, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum glucose, Follow-up, n=8, 9, 9 | 0.099 (0.3911) | 0.304 (0.5180) | 0.381 (0.3850)
  Serum calcium, Day 3 (48 hour), n=26, 26, 26 | 0.050 (0.0968) | 0.054 (0.0802) | 0.051 (0.0700)
  Serum calcium, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum calcium, Follow-up, n=8, 9, 9 | 0.003 (0.0861) | -0.019 (0.0692) | -0.046 (0.0865)
  Serum carbon dioxide, Day 3 (48 hour),n=26, 26, 26 | -0.2 (1.39) | -0.2 (1.22) | 0.0 (1.22)
  Serum carbon dioxide, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum carbon dioxide, Follow-up, n=8, 9, 9 | -1.4 (1.19) | -1.7 (1.58) | -1.6 (1.33)
  Serum chloride, Day 3 (48 hour),n=26, 26, 26 | -1.0 (1.78) | -1.1 (2.00) | -1.0 (2.27)
  Serum chloride, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum chloride, Follow-up, n=8, 9, 9 | 1.3 (1.75) | 0.7 (1.32) | 1.6 (2.24)
  Serum potassium, Day 3 (48 hour), n=26,26,26 | -0.06 (0.297) | -0.04 (0.270) | -0.06 (0.298)
  Serum potassium, Follow-up, n=8,9,9,: number analyzed (Participants) | 8 | 9 | 9
  Serum potassium, Follow-up, n=8,9,9, | -0.18 (0.306) | -0.09 (0.237) | -0.24 (0.371)
  Serum sodium, Day 3 (48 hour), n=26,26,26 | -0.3 (1.70) | -0.7 (1.67) | -0.5 (1.98)
  Serum sodium, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  Serum sodium, Follow-up, n=8,9,9 | -1.0 (2.39) | -1.3 (2.35) | -0.6 (1.74)
  Serum urea nitrogen, Day 3 (48 hour), n=26,26,26 | -0.250 (1.0929) | -0.307 (1.0021) | -0.332 (1.0598)
  Serum urea nitrogen, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  Serum urea nitrogen, Follow-up, n=8,9,9 | -0.043 (1.4732) | -0.354 (1.0294) | -0.223 (1.0126)

49. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Alanine Aminotransferase (ALT), Serum Alkaline Phosphatase (AP), Serum Aspartate Aminotransferase (AST) and Serum Creatinine Kinase (CK) for Part 1a
Description: Blood samples were collected for the assessment of chemistry parameters namely serum ALT, serum AP, serum AST and serum CK for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units/liter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
International units/liter
  Serum ALT, Day 3 (48 hour), n=26, 26, 26 | -1.1 (7.04) | -0.1 (7.30) | -0.3 (6.54)
  Serum ALT, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum ALT, Follow-up, n=8, 9, 9 | -3.0 (10.76) | 0.1 (11.57) | 5.4 (5.05)
  Serum AP, Day 3 (48 hour), n=26, 26, 26 | 7.7 (5.69) | 8.3 (5.40) | 9.0 (6.25)
  Serum AP, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum AP, Follow-up, n=8, 9, 9 | 2.6 (6.07) | 7.2 (7.71) | 7.4 (4.75)
  Serum AST, Day 3 (48 hour),n=26, 26, 26 | -0.6 (4.11) | -0.2 (4.01) | -0.5 (3.99)
  Serum AST, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum AST, Follow-up, n=8, 9, 9 | -0.1 (4.94) | 1.7 (7.18) | 3.1 (4.40)
  Serum CK, Day 3 (48 hour),n=26, 26, 26 | -28.7 (43.65) | -26.4 (47.32) | -30.2 (41.96)
  Serum CK, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum CK, Follow-up, n=8, 9, 9 | 8.0 (42.32) | 29.0 (107.27) | 13.2 (26.16)

50. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Albumin and Serum Protein for Part 1a
Description: Blood samples were collected for the assessment of chemistry parameters namely serum albumin and serum protein for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
grams/liter
  Serum albumin, Day 3 (48 hour), n=26, 26, 26 | 1.5 (2.27) | 1.8 (1.98) | 1.8 (2.36)
  Serum albumin, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum albumin, Follow-up, n=8, 9, 9 | -0.3 (2.55) | -0.7 (1.87) | -0.6 (2.46)
  Serum protein, Day 3 (48 hour), n=26, 26, 26 | 1.8 (4.68) | 1.9 (3.10) | 2.1 (3.98)
  Serum protein, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum protein, Follow-up, n=8, 9, 9 | -2.1 (4.29) | -2.6 (3.32) | -2.1 (4.43)

51. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Bilirubin, Serum Creatinine and Serum Direct Bilirubin for Part 1a
Description: Blood samples were collected for the assessment of chemistry parameters namely serum bilirubin, serum creatinine and serum direct bilirubin Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
micromoles/liter
  Serum bilirubin, Day 3 (48 hour), n=26, 26, 26 | 2.08 (2.746) | 1.59 (3.511) | 1.98 (3.018)
  Serum bilirubin, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum bilirubin, Follow-up, n=8, 9, 9 | 2.34 (3.608) | -1.08 (1.943) | -1.19 (4.431)
  Serum creatinine, Day 3 (48 hour), n=26, 26, 26 | 1.49 (5.758) | 2.14 (6.793) | 2.31 (6.564)
  Serum creatinine, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum creatinine, Follow-up, n=8, 9, 9 | 4.86 (5.349) | 2.28 (9.930) | 3.93 (5.859)
  Serum direct bilirubin, Day 3 (48 hour),n=26,26,26 | 0.25 (0.422) | 0.17 (0.528) | 0.18 (0.482)
  Serum direct bilirubin, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Serum direct bilirubin, Follow-up, n=8, 9, 9 | 0.46 (0.707) | -0.14 (0.384) | -0.09 (0.677)

52. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Basophils, Blood Eosinophils, Blood Leukocytes, Blood Lymphocytes, Blood Monocytes, Blood Neutrophils and Blood Platelets for Part 1a
Description: Blood samples were collected for the assessment of hematology parameters namely blood basophils, blood eosinophils, blood leukocytes, blood lymphocytes, blood monocytes, blood neutrophils and blood platelets for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
10^9 cells/liter
  Blood basophils, Day 3 (48 hour), n=26, 26, 26 | 0.004 (0.0344) | 0.004 (0.0344) | -0.004 (0.0344)
  Blood basophils, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood basophils, Follow-up, n=8, 9, 9 | 0.000 (0.0000) | 0.000 (0.0500) | 0.000 (0.0000)
  Blood eosinophils, Day 3 (48 hour), n=26, 26, 26 | 0.008 (0.0688) | 0.008 (0.0935) | 0.004 (0.0958)
  Blood eosinophils, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood eosinophils, Follow-up, n=8, 9, 9 | 0.025 (0.0463) | 0.044 (0.0527) | 0.033 (0.1323)
  Blood leukocytes, Day 3 (48 hour),n=26, 26, 26 | -0.388 (0.7464) | -0.300 (0.6957) | -0.400 (0.6675)
  Blood leukocytes, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood leukocytes, Follow-up, n=8, 9, 9 | -0.175 (0.4862) | 0.000 (1.2728) | -0.400 (0.3841)
  Blood lymphocytes, Day 3 (48 hour),n=26, 26, 26 | -0.050 (0.2832) | 0.015 (0.3081) | -0.008 (0.4127)
  Blood lymphocytes, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood lymphocytes, Follow-up, n=8, 9, 9 | 0.025 (0.2866) | -0.100 (0.4444) | 0.011 (0.2147)
  Blood monocytes, Day 3 (48 hour),n=26, 26, 26 | -0.065 (0.0977) | -0.069 (0.0970) | -0.096 (0.0871)
  Blood monocytes, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood monocytes, Follow-up, n=8, 9, 9 | 0.050 (0.0926) | 0.033 (0.1323) | -0.056 (0.0527)
  Blood neutrophils, Day 3 (48 hour),n=26, 26, 26 | -0.254 (0.5907) | -0.238 (0.5845) | -0.288 (0.4702)
  Blood neutrophils, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood neutrophils, Follow-up, n=8, 9, 9 | -0.213 (0.5330) | 0.089 (0.7976) | -0.356 (0.4187)
  Blood platelets, Day 3 (48 hour),n=26, 26, 26 | 11.5 (14.76) | 17.4 (16.43) | 14.5 (17.85)
  Blood platelets, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood platelets, Follow-up, n=8, 9, 9 | 3.8 (17.90) | 1.8 (17.89) | 9.8 (26.48)

53. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Erythrocyte (Ery.) Mean Corpuscular Hemoglobin Concentration (MCHC) and Blood Hemoglobin for Part 1a
Description: Blood samples were collected for the assessment of hematology parameters namely blood Ery. MCHC and blood hemoglobin for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
grams/liter
  Blood Ery. MCHC, Day 3 (48 hour), n=26, 26, 26 | 0.4 (4.78) | 0.9 (4.27) | 0.4 (5.56)
  Blood Ery. MCHC, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood Ery. MCHC, Follow-up, n=8, 9, 9 | 2.5 (6.63) | 4.1 (3.33) | 3.0 (5.52)
  Blood hemoglobin, Day 3 (48 hour), n=26, 26, 26 | 8.0 (7.21) | 8.5 (6.59) | 8.4 (7.26)
  Blood hemoglobin, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood hemoglobin, Follow-up, n=8, 9, 9 | -3.8 (6.45) | -4.4 (6.29) | -2.3 (8.03)

54. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. Mean Corpuscular Hemoglobin (MCH) for Part 1a
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCH for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
picograms
  Blood Ery.MCH, Day 3 (48 hour), n=26, 26, 26 | -0.03 (0.360) | 0.00 (0.280) | -0.02 (0.400)
  Blood Ery. MCH, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood Ery. MCH, Follow-up, n=8, 9, 9 | -0.03 (0.512) | 0.14 (0.270) | 0.04 (0.317)

55. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. Mean Corpuscular Volume (MCV) for Part 1a
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCV for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
femtoliters
  Blood Ery. MCV, Day 3 (48 hour), n=26, 26, 26 | -0.21 (0.471) | -0.26 (0.568) | -0.23 (0.586)
  Blood Ery. MCV, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood Ery. MCV, Follow-up, n=8, 9, 9 | -0.73 (0.618) | -0.58 (0.549) | -0.72 (0.800)

56. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. for Part 1a
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
10^12 cells/liter
  Blood Ery. , Day 3 (48 hour), n=26, 26, 26 | 0.279 (0.2597) | 0.293 (0.2450) | 0.296 (0.2538)
  Blood Ery. , Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood Ery. , Follow-up, n=8, 9, 9 | -0.130 (0.2045) | -0.190 (0.2258) | -0.101 (0.2538)

57. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hematocrit for Part 1a
Description: Blood samples were collected for the assessment of hematology parameter namely blood hematocrit for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
Percentage of red blood cells in blood
  Blood hematocrit , Day 3 (48 hour), n=26, 26, 26 | 2.32 (2.212) | 2.43 (2.110) | 2.48 (2.200)
  Blood hematocrit, Follow-up, n=8, 9, 9: number analyzed (Participants) | 8 | 9 | 9
  Blood hematocrit, Follow-up, n=8, 9, 9 | -1.50 (1.628) | -1.87 (1.781) | -1.20 (2.029)

58. Secondary Outcome: Change From Baseline in Vital Sign Parameters Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) for Part 1a
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included SBP, DBP. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety population
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
millimeters of mercury
  SBP, Day 1 (2 hours), n=26, 26, 26, | 1.8 (6.88) | -1.3 (7.24) | 1.1 (5.25)
  SBP, Day 2 (24 hours), n=26, 26, 26 | 0.1 (6.82) | -2.8 (10.21) | -1.8 (5.31)
  SBP, Day 3 (48 hours), n=26, 26, 26 | 5.3 (7.93) | -1.3 (7.12) | -0.2 (6.46)
  SBP, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  SBP, Follow-up, n=8,9,9 | 18.0 (11.28) | 9.4 (6.09) | 6.9 (7.83)
  DBP, Day 1 (2 hours), n=26, 26, 26, | 3.2 (7.04) | 1.0 (5.59) | 2.2 (6.34)
  DBP, Day 2 (24 hours), n=26, 26, 26 | 2.3 (8.11) | -0.4 (7.41) | 0.0 (6.87)
  DBP, Day 3 (48 hours), n=26, 26, 26 | 2.2 (7.65) | 2.8 (6.29) | 1.0 (7.19)
  DBP, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  DBP, Follow-up, n=8,9,9 | 8.3 (7.36) | 6.4 (5.73) | 7.4 (4.85)

59. Secondary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part 1a
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
beats/minute
  Heart rate, Day 1 (2 hours), n=26, 26, 26, | -0.7 (7.59) | 0.0 (4.61) | 1.7 (3.61)
  Heart rate, Day 2 (24 hours), n=26, 26, 26 | -0.7 (7.11) | 0.6 (5.87) | 1.7 (3.82)
  Heart rate, Day 3 (48 hours), n=26, 26, 26 | -0.2 (8.18) | -0.2 (6.20) | 3.2 (5.46)
  Heart rate, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  Heart rate, Follow-up, n=8,9,9 | -0.1 (3.04) | 0.2 (7.56) | 5.7 (5.15)

60. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter Heart Rate for Part 1a
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that automatically calculated the heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
beats per minute
  ECG Heart rate, Day 1 (2 hours), n=26, 26, 26, | -1.1 (6.33) | -1.0 (6.05) | 0.4 (3.60)
  ECG Heart rate, Day 2 (24 hours), n=26, 26, 26 | 0.2 (5.85) | -0.4 (8.02) | 0.3 (3.96)
  ECG Heart rate, Day 3 (48 hours), n=26, 26, 26 | 0.0 (6.39) | -0.6 (7.00) | 1.0 (4.04)
  ECG Heart rate, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  ECG Heart rate, Follow-up, n=8,9,9 | -1.0 (4.11) | 0.7 (8.82) | 3.6 (6.56)

61. Secondary Outcome: Change From Baseline in ECG Parameters PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Bazett's Formula (QTcB) and Corrected QT Interval Using Fridericia's Formula (QTcF) for Part 1a
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that measured PR interval, QRS duration, QT interval, QTcB and QTcF for Part 1a. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
milliseconds
  PR interval, Day 1 (2 hours), n=26, 26, 26 | -2.5 (12.28) | -3.2 (11.79) | -3.8 (6.01)
  PR interval, Day 2 (24 hours), n=26, 26, 26 | 1.7 (13.77) | -0.1 (8.80) | -0.5 (9.20)
  PR interval,, Day 3 (48 hours), n=26, 26, 26 | 1.2 (9.64) | -0.3 (7.74) | 2.0 (12.51)
  PR interval, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  PR interval, Follow-up, n=8,9,9 | 4.0 (14.89) | -3.1 (9.98) | -9.2 (7.41)
  QRS duration, Day 1 (2 hours), n=26, 26, 26, | 1.3 (4.65) | 0.1 (5.61) | -0.4 (4.64)
  QRS duration, Day 2 (24 hours), n=26, 26, 26 | 0.3 (3.64) | -1.0 (5.62) | -0.5 (5.07)
  QRS duration, Day 3 (48 hours), n=26, 26, 26 | 0.1 (4.47) | -0.1 (5.42) | -1.8 (5.28)
  QRS duration, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  QRS duration, Follow-up, n=8,9,9 | -0.4 (7.21) | 2.1 (8.31) | 0.9 (2.26)
  QT interval Day 1 (2 hours), n=26, 26, 26, | 9.6 (14.42) | 6.4 (12.07) | 8.8 (11.28)
  QT interval, Day 2 (24 hours), n=26, 26, 26 | 1.5 (11.55) | 2.1 (15.22) | 2.4 (8.40)
  QT interval, Day 3 (48 hours), n=26, 26, 26 | 1.8 (12.95) | -0.5 (14.55) | -0.7 (10.80)
  QT interval, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  QT interval, Follow-up, n=8,9,9 | 17.5 (22.99) | 5.2 (29.79) | -3.6 (17.81)
  QTcB interval, Day 1 (2 hours), n=26, 26, 26, | 6.6 (14.07) | 4.3 (14.96) | 10.3 (11.26)
  QTcB, Day 2 (24 hours), n=26, 26, 26 | 1.8 (12.63) | 1.7 (13.74) | 3.8 (9.86)
  QTcB, Day 3 (48 hours), n=26, 26, 26 | 2.0 (12.56) | -1.6 (13.26) | 2.9 (9.76)
  QTcB, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  QTcB, Follow-up, n=8,9,9 | 13.9 (19.95) | 2.9 (19.62) | 6.0 (11.51)
  QTcF interval, Day 1 (2 hours), n=26, 26, 26, | 7.5 (10.56) | 4.8 (11.05) | 10.0 (9.57)
  QTcF, Day 2 (24 hours), n=26, 26, 26 | 1.7 (9.11) | 2.0 (9.73) | 3.4 (7.21)
  QTcF, Day 3 (48 hours), n=26, 26, 26 | 2.0 (8.30) | -1.3 (9.93) | 1.8 (8.20)
  QTcF, Follow-up, n=8,9,9: number analyzed (Participants) | 8 | 9 | 9
  QTcF, Follow-up, n=8,9,9 | 15.4 (20.16) | 4.9 (18.84) | 4.6 (7.65)

62. Secondary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Analysis Part 1a
Description: Urinalysis parameters assessed were urine ketones, urine glucose, urine occult blood, urine pH, urine specific gravity and urine protein. In this dipstick test, the level of ketones, glucose, occult blood, pH, specific gravity and protein in urine samples was recorded as negative trace, 1+, 3+, 5+, 6+, 7+ and 8+ (the plus sign increases with a higher level of ketones, occult blood, pH or specific gravity in the urine: 1+=slightly positive, 3+ to 5+=positive, 6+ and above=high positive). Urine samples were collected for the measurement of urinalysis parameters by dipstick method up-to follow-up (5 to 7 days post last dose) in Part 1a. Only categories with significant values have been presented.
Time Frame: Up to 14 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets
Number analyzed (Participants) | 26 | 26 | 26
Participants
  Urine Ketones, Day 3 (48 hours), 1+ | 1 | 0 | 0
  Urine pH, Day 3 (48 hours), 5+ | 4 | 4 | 4
  Urine pH, Day 3 (48 hours), 6+ | 18 | 16 | 14
  Urine pH, Day 3 (48 hours), 7+ | 3 | 6 | 8
  Urine pH, Day 3 (48 hours), 8+ | 1 | 0 | 0
  Urine pH, Follow-up, 5+ | 2 | 4 | 3
  Urine pH, Follow-up, 6+ | 5 | 5 | 4
  Urine pH, Follow-up, 7+ | 1 | 0 | 2
  Urine Specific gravity, Day 3 (48 hours), 1+ | 26 | 26 | 26
  Urine Specific gravity, Follow-up, 1+ | 8 | 9 | 9

63. Secondary Outcome: Number of Participants With AEs and SAEs for Part 1b
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Up to 11 days
Population: Safety Population. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Glucose, Serum Calcium, Serum Carbon Dioxide, Serum Chloride, Serum Potassium, Serum Sodium and Serum Urea Nitrogen for Part 1b
Description: Blood samples were collected for the assessment of chemistry parameters namely serum glucose, serum calcium, serum carbon dioxide, serum chloride, serum potassium, serum sodium and serum urea nitrogen for Part 1b. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

65. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum ALT, Serum AP, Serum AST and Serum CK for Part 1b
Description: Blood samples were collected for the assessment of chemistry parameters namely serum ALT, serum AP, serum AST and serum CK for Part 1b. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

66. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Albumin and Serum Protein for Part 1b
Description: Blood samples were collected for the assessment of chemistry parameters namely serum albuim and serum protein for Part 1b. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

67. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Bilirubin, Serum Creatinine and Serum Direct Bilirubin in Part 1b
Description: as for outcome 65
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

68. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Basophils, Blood Eosinophils, Blood Leukocytes, Blood Lymphocytes, Blood Monocytes, Blood Neutrophils and Blood Platelets for Part 1b
Description: Blood samples were collected for the assessment of hematology parameters namely blood basophils, blood eosinophils, blood leukocytes, blood lymphocytes, blood monocytes, blood neutrophils and blood platelets for Part 1b. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

69. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Ery. MCHC and Blood Hemoglobin for Part 1b
Description: Blood samples were collected for the assessment of hematology parameters namely blood Ery. MCHC and blood hemoglobin for Part 1b. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

70. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. MCH for Part 1b
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCH for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

71. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. MCV for Part 1b
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCV for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Groups:
- Gepotidacin 3000 mg RC Tablets-fed: Participants received Gepotidacin 1500 mg (2 x 750 mg) RC tablets orally in the fed state in one of the 2 treatment periods for 3 days in Part 1a.
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

72. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. for Part 1b
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. for Part 1b. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

73. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hematocrit for Part 1b
Description: Blood samples were collected for the assessment of hematology parameter namely blood hematocrit for Part 1b. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

74. Secondary Outcome: Change From Baseline in Vital Sign Parameters SBP and DBP for Part 1b
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included SBP, DBP. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

75. Secondary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part 1b
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

76. Secondary Outcome: Change From Baseline in ECG Parameter Heart Rate for Part 1b
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that automatically calculated the heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

77. Secondary Outcome: Change From Baseline in ECG Parameters PR Interval, QRS Duration, QT Interval, QTcB and QTcF for Part 1b
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that measured PR interval, QRS duration, QT interval, QTcB and QTcF for Part 1b. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Baseline and up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

78. Secondary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Analysis Part 1b
Description: Urinalysis parameters assessed were urine ketones, urine glucose, urine occult blood, urine pH, urine specific gravity and urine protein. In this dipstick test, the level of ketones, glucose, occult blood, pH, specific gravity and protein in urine samples was recorded as negative trace, 1+, 3+, 5+, 6+, 7+ and 8+ (the plus sign increases with a higher level of ketones, occult blood, pH or specific gravity in the urine: 1+=slightly positive, 3+ to 5+=positive, 6+ and above=high positive). Since the relative bio-availability of the RC tablet formulation under fasted and fed conditions had been previously evaluated in Study BTZ117349 (NCT02045849), Part 1b was not conducted.
Time Frame: Up to 11 days
Population: as for outcome 63
Arm/Group | Gepotidacin 1500 mg RC Tablets-fasted | Gepotidacin 3000 mg RC Tablets-fed
Number analyzed (Participants) | 0 | 0

79. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs for Part 2
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 11 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
Participants
  Non serious AE | 6 | 9
  SAE | 0 | 0

80. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Glucose, Serum Calcium, Serum Carbon Dioxide, Serum Chloride, Serum Potassium, Serum Sodium and Serum Urea Nitrogen in Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely serum glucose, serum calcium, serum carbon dioxide, serum chloride, serum potassium, serum sodium and serum urea nitrogen for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
millimoles/liter
  Serum glucose, Day 3 (48 hour) | -0.146 (0.4421) | -0.133 (0.3665)
  Serum glucose, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.211 (0.5005)
  Serum calcium, Day 3 (48 hour) | -0.027 (0.1055) | -0.009 (0.0684)
  Serum calcium, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.011 (0.0638)
  Serum carbon dioxide, Day 3 (48 hour) | 1.5 (1.96) | -1.4 (1.71)
  Serum carbon dioxide, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.4 (1.78)
  Serum chloride, Day 3 (48 hour) | -1.5 (1.96) | -1.2 (2.04)
  Serum chloride, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 0.1 (2.13)
  Serum potassium, Day 3 (48 hour) | -0.03 (0.437) | -0.16 (0.517)
  Serum potassium, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 0.01 (0.446)
  Serum sodium, Day 3 (48 hour) | -1.1 (1.45) | -0.9 (2.02)
  Serum sodium, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 0.4 (2.22)
  Serum urea nitrogen, Day 3 (48 hour) | 0.678 (0.8489) | 1.321 (1.2692)
  Serum urea nitrogen, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 0.216 (1.7478)

81. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum ALT, Serum AP, Serum AST and Serum CK in Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely serum ALT, serum AP, serum AST and serum CK for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
International units/liter
  Serum ALT, Day 3 (48 hour) | -0.2 (1.55) | 1.3 (3.16)
  Serum ALT, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 3.1 (5.95)
  Serum AP, Day 3 (48 hour) | -0.3 (5.44) | -0.3 (4.00)
  Serum AP, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -1.7 (2.95)
  Serum AST, Day 3 (48 hour) | 0.5 (2.92) | 1.0 (2.71)
  Serum AST, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 3.5 (4.81)
  Serum CK, Day 3 (48 hour) | -22.7 (26.45) | -25.7 (15.81)
  Serum CK, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -9.8 (13.99)

82. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Albumin and Serum Protein for Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely serum albumin and serum protein for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
grams/liter
  Serum albumin, Day 3 (48 hour) | -0.9 (3.38) | 0.0 (1.70)
  Serum albumin, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -1.5 (2.17)
  Serum protein, Day 3 (48 hour) | 0.0 (5.29) | -2.1 (4.63)
  Serum protein, Follow-up, | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -1.8 (2.70)

83. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Bilirubin, Serum Creatinine and Serum Direct Bilirubin for Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely serum bilirubin, serum creatinine and serum direct bilirubin for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
micromoles/liter
  Serum bilirubin, Day 3 (48 hour) | -1.02 (2.944) | -3.62 (2.968)
  Serum bilirubin | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.68 (4.207)
  Serum creatinine, Day 3 (48 hour) | -1.76 (8.147) | -4.42 (6.254)
  Serum creatinine | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -3.55 (7.458)
  Serum direct bilirubin, Day 3 (48 hour) | -0.51 (1.147) | -1.02 (0.878)
  Serum direct bilirubin, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.34 (1.075)

84. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter Serum Estradiol for Part 2
Description: Blood samples were collected for the assessment of chemistry parameter namely serum estradiol for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the indicated time point were analyzed. NA indicates standard deviation was not calculated as a single participant was analyzed.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: picomoles/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 1 | 1
picomoles/liter | NA (NA) — Standard deviation was not calculated as a single participant was analyzed. | 0.00 (NA) — Standard deviation was not calculated as a single participant was analyzed.

85. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Basophils, Blood Eosinophils, Blood Leukocytes, Blood Lymphocytes, Blood Monocytes, Blood Neutrophils and Blood Platelets for Part 2
Description: Blood samples were collected for the assessment of hematology parameters namely blood basophils, blood eosinophils, blood leukocytes, blood lymphocytes, blood monocytes, blood neutrophils and blood platelets for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
10^9 cells/liter
  Blood basophils, Day 3 (48 hour) | 0.002 (0.0092) | 0.009 (0.0129)
  Blood basophils, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 0.004 (0.0097)
  Blood eosinophils, Day 3 (48 hour) | 0.036 (0.0626) | 0.052 (0.0839)
  Blood eosinophils, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 0.021 (0.0671)
  Blood leukocytes, Day 3 (48 hour) | 0.129 (0.7779) | 0.039 (0.8843)
  Blood leukocytes, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.183 (0.7906)
  Blood lymphocytes, Day 3 (48 hour) | 0.222 (0.1707) | 0.243 (0.2165)
  Blood lymphocytes, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.038 (0.2875)
  Blood monocytes, Day 3 (48 hour) | -0.020 (0.0651) | -0.013 (0.0732)
  Blood monocytes, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 0.045 (0.0546)
  Blood neutrophils, Day 3 (48 hour) | -0.112 (0.6906) | -0.251 (0.6701)
  Blood neutrophils, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.213 (0.8126)
  Blood platelets, Day 3 (48 hour) | -7.4 (38.14) | -0.6 (33.37)
  Blood platelets, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 2.1 (31.49)

86. Secondary Outcome: Change From Baseline in Hematology Parameters Ery. MCHC and Blood Hemoglobin for Part 2
Description: Blood samples were collected for the assessment of hematology parameters namely blood Ery. MCHC and blood hemoglobin for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
grams/liter
  Blood Ery. MCHC, Day 3 (48 hour) | -6.6 (4.35) | -6.6 (3.20)
  Blood Ery. MCHC, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2 | -6.2 (5.87)
  Blood hemoglobin, Day 3 (48 hour) | 2.8 (9.43) | 0.9 (5.55)
  Blood hemoglobin, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2 | -5.9 (3.67)

87. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. MCH for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCH for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
picograms
  Blood Ery.MCH, Day 3 (48 hour) | -0.25 (0.331) | -0.06 (0.378)
  Blood Ery. MCH, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.15 (0.488)

88. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. MCV for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCV for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
femtoliters
  Blood Ery. MCV, Day 3 (48 hour) | 1.17 (1.610) | 1.69 (1.371)
  Blood Ery. MCV, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 1.28 (1.834)

89. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
10^12 cells/liter
  Blood Ery., Day 3 (48 hour) | 0.118 (0.2839) | 0.033 (0.1675)
  Blood Ery., Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.175 (0.1099)

90. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hematocrit for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely blood hematocrit for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
Percentage of red blood cells in blood
  Blood hematocrit , Day 3 (48 hour) | 1.6 (2.871) | 1.02 (1.713)
  Blood hematocrit, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -1.09 (1.079)

91. Secondary Outcome: Change From Baseline in Vital Sign Parameters SBP and DBP for Part 2
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included SBP, DBP. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety population
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
millimeters of mercury
  SBP, Day 1 (2 hours) | -8.4 (15.78) | 6.7 (10.49)
  SBP, Day 2 (24 hours) | -9.6 (13.55) | -3.1 (12.90)
  SBP, Day 3 (48 hours) | -4.1 (17.99) | -4.2 (11.03)
  SBP, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -2.0 (17.81)
  DBP, Day 1 (2 hours) | -6.7 (6.13) | -0.3 (6.95)
  DBP, Day 2 (24 hours) | -5.4 (8.72) | -3.5 (6.92)
  DBP, Day 3 (48 hours) | -1.9 (7.98) | -1.7 (6.62)
  DBP, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -0.1 (11.35)

92. Secondary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part 2
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
beats/minute
  Heart rate, Day 1 (2 hours) | 0.1 (7.84) | 3.2 (6.48)
  Heart rate, Day 2 (24 hours) | -3.8 (12.38) | -1.4 (6.90)
  Heart rate, Day 3 (48 hours) | -3.0 (11.22) | 3.4 (6.29)
  Heart rate, Follow-up | NA (NA) — NA indicates participants crossed-over as follow-up visit occurred after Period 2. | -0.3 (9.06)

93. Secondary Outcome: Change From Baseline in ECG Parameter Heart Rate for Part 2
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that automatically calculated the heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
beats/minute
  ECG Heart rate, Day 1 (2 hours) | 5.4 (10.13) | 4.9 (5.02)
  ECG Heart rate, Day 2 (24 hours) | -1.2 (8.75) | -1.1 (6.71)
  ECG Heart rate, Day 3 (48 hours) | 2.1 (11.00) | 3.4 (5.38)
  ECG Heart rate, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -1.6 (8.18)

94. Secondary Outcome: Change From Baseline in ECG Parameters PR Interval, QRS Duration, QT Interval, QTcB and QTcF for Part 2
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that measured PR interval, QRS duration, QT interval, QTcB and QTcF for Part 2. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. NA indicates participants crossed-over as follow-up visit occurred after Period 2.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
milliseconds
  PR interval, Day 1 (2 hours) | -1.7 (13.92) | 0.5 (11.49)
  PR interval, Day 2 (24 hours) | 7.2 (11.44) | -2.7 (7.23)
  PR interval, Day 3 (48 hours) | 5.1 (11.46) | 3.0 (11.71)
  PR interval, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | -1.2 (15.37)
  QRS duration, Day 1 (2 hours) | 0.4 (5.19) | 3.9 (4.28)
  QRS duration, Day 2 (24 hours) | 0.3 (4.57) | -0.2 (4.73)
  QRS duration, Day 3 (48 hours) | -0.2 (4.54) | 0.7 (4.06)
  QRS duration, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 1.6 (3.60)
  QT interval Day 1 (2 hours) | -4.0 (16.21) | 5.1 (16.04)
  QT interval, Day 2 (24 hours) | 4.8 (21.63) | 11.7 (17.31)
  QT interval, Day 3 (48 hours) | -1.0 (20.48) | -3.4 (14.95)
  QT interval, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 9.5 (17.37)
  QTcB interval, Day 1 (2 hours) | 15.2 (18.23) | 20.7 (14.17)
  QTcB, Day 2 (24 hours) | 3.4 (11.64) | 9.5 (8.24)
  QTcB, Day 3 (48 hours) | 6.6 (16.26) | 6.0 (13.00)
  QTcB, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 5.7 (13.44)
  QTcF interval, Day 1 (2 hours) | 8.6 (9.56) | 15.2 (13.09)
  QTcF, Day 2 (24 hours) | 4.0 (10.23) | 10.4 (8.75)
  QTcF, Day 3 (48 hours) | 4.0 (8.60) | 2.4 (11.64)
  QTcF, Follow-up | NA (NA) — Participants crossed-over as follow-up visit occurred after Period 2. | 7.0 (9.36)

95. Secondary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Analysis Part 2
Description: Urinalysis parameters assessed were urine ketones, urine glucose, urine occult blood, urine pH, urine specific gravity and urine protein. In this dipstick test, the level of ketones, glucose, occult blood, pH, specific gravity and protein in urine samples was recorded as negative trace, 1+, 3+, 4+ 5+, 6+, 7+ and 8+ (the plus sign increases with a higher level of ketones, occult blood, pH or specific gravity in the urine: 1+=slightly positive, 3+ to 5+=positive, 6+ and above=high positive). Urine samples were collected for the measurement of urinalysis parameters by dipstick method up-to follow-up (5 to 7 days post last dose) in Part 2. Only categories with significant values have been presented.
Time Frame: Baseline and up to 11 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets
Number analyzed (Participants) | 10 | 10
Participants
  Urine Ketones, Follow-up, Trace | 0 | 1
  Urine Occult blood, Day 3 (48 hours), 1+ | 0 | 1
  Urine Occult blood, Trace, Day 3 (48 hours), | 2 | 0
  Urine Occult blood, Follow-up, 1+ | 0 | 1
  Urine pH, Day 3 (48 hours), 5+ | 2 | 7
  Urine pH, Day 3 (48 hours), 6+ | 6 | 2
  Urine pH, Day 3 (48 hours), 7+ | 1 | 1
  Urine pH, Day 3 (48 hours), 8+ | 1 | 0
  Urine pH, Follow-up, 5+ | 0 | 3
  Urine pH, Follow-up, 6+ | 0 | 6
  Urine pH, Follow-up, 8+ | 0 | 1
  Urine Specific gravity, Day 3 (48 hours), 1+ | 10 | 10
  Urine Specific gravity, Follow-up, 1+ | 0 | 10

96. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs for Part 3
Description: as for outcome 79
Time Frame: Up to 14 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Gepotidacin RC 1500 mg Fed: Participants received a single dose gepotidacin 1500mg (2 x 750 mg) RC tablets in the fed state orally in Part 3 Period 1.
- Gepotidacin RC 2250 mg Fed: Participants received a single dose gepotidacin 2250mg (3 x 750 mg) RC tablets in the fed state orally in Part 3 Period 2.
- Gepotidacin RC 3000 mg Fed: Participants received a single dose gepotidacin 3000mg (4 x 750 mg) RC tablets in the fed state orally in Part 3 Period 3.
- Placebo: Participants received matching placebo to active tablets in the fed state in one of the 3 treatment periods in Part 3.
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
Participants
  Non seriou AE | 0 | 1 | 6 | 0
  SAE | 0 | 0 | 0 | 0

97. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Glucose, Serum Calcium, Serum Carbon Dioxide, Serum Chloride, Serum Potassium, Serum Sodium and Serum Urea Nitrogen for Part 3
Description: Blood samples were collected for the assessment of chemistry parameters namely serum glucose, serum calcium, serum carbon dioxide, serum chloride, serum potassium, serum sodium and serum urea nitrogen for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
millimoles/liter
  Glucose,Period 1,Day 3(48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Glucose,Period 1,Day 3(48 hour),n=10,0,0,2 | 0.038 (0.3178) |  |  | -0.305 (0.4313)
  Glucose,Period 2,Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Glucose,Period 2,Day 3 (48 hour),n=0,10,0,2 |  | -0.071 (0.2993) |  | -0.415 (0.2758)
  Glucose,Period 3,Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Glucose,Period 3,Day 3 (48 hour),n=0,0,9,2 |  |  | -0.197 (0.2355) | -0.335 (0.1626)
  Glucose, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Glucose, Follow-up, n=0,0,9,2 |  |  | -0.050 (0.2744) | -0.390 (0.3960)
  Calcium,Period1, Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Calcium,Period1, Day 3 (48 hour),n=10,0,0,2 | -0.057 (0.0887) |  |  | -0.075 (0.1061)
  Calcium,Period 2,Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Calcium,Period 2,Day 3 (48 hour),n=0,10,0,2 |  | -0.046 (0.0819) |  | -0.115 (0.0919)
  Calcium,Period 3,Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Calcium,Period 3,Day 3 (48 hour),n=0,0,9,2 |  |  | -0.028 (0.0502) | -0.105 (0.0354)
  Calcium, Follow-up, n=0,0, 9, 2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Calcium, Follow-up, n=0,0, 9, 2 |  |  | -0.039 (0.0742) | -0.040 (0.0141)
  Carbon dioxide,Period 1,Day 3(48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Carbon dioxide,Period 1,Day 3(48 hour),n=10,0,0,2 | -0.6 (1.51) |  |  | 0.5 (0.71)
  Carbon dioxide,Period 2,Day 3(48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Carbon dioxide,Period 2,Day 3(48 hour),n=0,10,0,2 |  | -0.7 (1.64) |  | 2.5 (2.12)
  Carbon dioxide,Period 3,Day 3(48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Carbon dioxide,Period 3,Day 3(48 hour),n=0,0,9,2 |  |  | -1.1 (1.36) | 1.5 (0.71)
  Carbon dioxide, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Carbon dioxide, Follow-up, n=0,0,9,2 |  |  | 0.2 (2.28) | 1.5 (0.71)
  Chloride, Period 1, Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Chloride, Period 1, Day 3 (48 hour),n=10,0,0,2 | 0.8 (1.23) |  |  | 1.0 (2.83)
  Chloride, Period 2, Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Chloride, Period 2, Day 3 (48 hour),n=0,10,0,2 |  | 0.8 (1.75) |  | -2.0 (0.00)
  Chloride, Period 3, Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Chloride, Period 3, Day 3 (48 hour),n=0,0,9,2 |  |  | 0.1 (1.96) | -1.5 (0.71)
  Chloride, Follow-up,n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Chloride, Follow-up,n=0,0,9,2 |  |  | 0.2 (2.95) | -2.0 (0.00)
  Potassium, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Potassium, Period 1, Day 3 (48 hour), n=10,0,0,2 | -0.21 (0.536) |  |  | -0.10 (0.283)
  Potassium, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Potassium, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | -0.19 (0.381) |  | -0.40 (1.131)
  Potassium, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Potassium, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | -0.28 (0.561) | -0.30 (1.273)
  Potassium, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Potassium, Follow-up, n=0,0,9,2 |  |  | -0.21 (0.359) | -0.15 (0.919)
  Sodium, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Sodium, Period 1, Day 3 (48 hour), n=10,0,0,2 | 0.6 (2.12) |  |  | 2.5 (2.12)
  Sodium, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Sodium, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | 0.1 (2.38) |  | -1.0 (2.83)
  Sodium, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Sodium, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | 0.3 (1.94) | -2.0 (4.24)
  Sodium, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Sodium, Follow-up, n=0,0,9,2 |  |  | -0.1 (1.90) | -2.5 (2.12)
  Urea nitrogen,Period 1,Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Urea nitrogen,Period 1,Day 3 (48 hour),n=10,0,0,2 | 0.606 (1.0760) |  |  | 0.535 (0.2475)
  Urea nitrogen,Period 2,Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Urea nitrogen,Period 2,Day 3 (48 hour),n=0,10,0,2 |  | 0.677 (1.3401) |  | 1.610 (0.7637)
  Urea nitrogen,Period 3,Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Urea nitrogen,Period 3,Day 3 (48 hour),n=0,0,9,2 |  |  | 0.474 (1.4617) | 1.075 (0.0071)
  Urea nitrogen, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Urea nitrogen, Follow-up, n=0,0,9,2 |  |  | 0.356 (1.2998) | 2.320 (2.7860)

98. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum ALT, Serum AP, Serum AST and Serum CK for Part 3
Description: Blood samples were collected for the assessment of chemistry parameters namely serum ALT, serum AP, serum AST and serum CK for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units/liter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
International units/liter
  ALT, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  ALT, Period 1, Day 3 (48 hour), n=10,0,0,2 | 0.1 (2.73) |  |  | -2.5 (2.12)
  ALT, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  ALT, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | 2.2 (3.36) |  | -4.0 (7.07)
  ALT, Period 3, Day 3 (48 hour), n=0,0,9,2,: number analyzed (Participants) | 0 | 0 | 9 | 2
  ALT, Period 3, Day 3 (48 hour), n=0,0,9,2, |  |  | 6.0 (3.74) | -4.5 (9.19)
  ALT, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  ALT, Follow-up, n=0,0,9,2 |  |  | 5.9 (4.11) | -5.0 (11.31)
  AP, Period 1, Day 3 (48 hour), n=10,0,0,2,: number analyzed (Participants) | 10 | 0 | 0 | 2
  AP, Period 1, Day 3 (48 hour), n=10,0,0,2, | -3.6 (2.07) |  |  | -9.0 (5.66)
  AP, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  AP, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | -2.5 (4.62) |  | -2.0 (4.24)
  Serum AP, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Serum AP, Day 3 (48 hour), n=0,0,9,2 |  |  | 0.6 (3.88) | -0.5 (0.71)
  AP, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  AP, Follow-up, n=0,0,9,2 |  |  | 1.8 (3.96) | 3.5 (3.54)
  AST, Period 1, Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  AST, Period 1, Day 3 (48 hour),n=10,0,0,2 | 1.3 (3.06) |  |  | -3.5 (2.12)
  AST, Period 2, Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  AST, Period 2, Day 3 (48 hour),n=0,10,0,2 |  | 1.7 (2.50) |  | -5.0 (4.24)
  AST, Period 3, Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  AST, Period 3, Day 3 (48 hour),n=0,0,9,2 |  |  | 4.2 (2.68) | -5.0 (5.66)
  AST, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  AST, Follow-up, n=0,0,9,2 |  |  | 2.6 (2.46) | -4.0 (7.07)
  CK, Period 1, Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  CK, Period 1, Day 3 (48 hour),n=10,0,0,2 | -28.1 (17.60) |  |  | -22.5 (14.85)
  CK, Period 2, Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  CK, Period 2, Day 3 (48 hour),n=0,10,0,2 |  | -11.8 (65.84) |  | -33.5 (23.33)
  CK, Period 3, Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  CK, Period 3, Day 3 (48 hour),n=0,0,9,2 |  |  | -14.3 (20.27) | -21.5 (9.19)
  CK, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  CK, Follow-up, n=0,0,9,2 |  |  | 3.7 (26.87) | 1.0 (11.31)

99. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Albumin and Serum Protein for Part 3
Description: Blood samples were collected for the assessment of chemistry parameters namely serum albumin and serum protein for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
grams/liter
  Albumin, Part 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Albumin, Part 1, Day 3 (48 hour), n=10,0,0,2 | -2.0 (2.54) |  |  | -2.0 (0.00)
  Albumin, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Albumin, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | -2.0 (1.05) |  | -3.0 (1.41)
  Albumin, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Albumin, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | -0.6 (3.05) | -2.5 (0.71)
  Albumin, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Albumin, Follow-up, n=0,0,9,2 |  |  | -0.3 (3.12) | -0.5 (2.12)
  Protein, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Protein, Period 1, Day 3 (48 hour), n=10,0,0,2 | -3.0 (2.31) |  |  | -4.5 (0.71)
  Protein, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Protein, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | -2.2 (3.01) |  | -5.0 (1.41)
  Protein, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Protein, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | -0.6 (3.97) | -4.5 (0.71)
  Protein, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Protein, Follow-up, n=0,0,9,2 |  |  | -0.6 (4.64) | -1.0 (5.66)

100. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Serum Bilirubin and Serum Creatinine for Part 3
Description: Blood samples were collected for the assessment of chemistry parameters namely serum bilirubin and serum creatinine for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
micromoles/liter
  Bilirubin, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Bilirubin, Period 1, Day 3 (48 hour), n=10,0,0,2 | -2.43 (3.364) |  |  | -0.85 (1.202)
  Bilirubin, Period 2, Day 3 (48 hour), n=0,10,0,2,: number analyzed (Participants) | 0 | 10 | 0 | 2
  Bilirubin, Period 2, Day 3 (48 hour), n=0,10,0,2, |  | -3.11 (3.793) |  | -1.70 (0.000)
  Bilirubin, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Bilirubin, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | -2.28 (3.844) | 0.85 (1.202)
  Bilirubin, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Bilirubin, Follow-up, n=0,0,9,2 |  |  | -1.53 (2.757) | -1.70 (0.000)
  Creatinine, Period 1,Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Creatinine, Period 1,Day 3 (48 hour), n=10,0,0,2 | -1.75 (8.101) |  |  | -17.65 (12.516)
  Creatinine, Period 2,Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Creatinine, Period 2,Day 3 (48 hour), n=0,10,0,2 |  | -1.75 (6.958) |  | -17.60 (0.000)
  Creatinine, Period 3,Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Creatinine, Period 3,Day 3 (48 hour), n=0,0,9,2 |  |  | 0.01 (7.636) | -13.20 (6.223)
  Creatinine, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Creatinine, Follow-up, n=0,0,9,2 |  |  | 2.97 (6.258) | -4.40 (6.223)

101. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Basophils, Blood Eosinophils, Blood Leukocytes, Blood Lymphocytes, Blood Monocytes, Blood Neutrophils and Blood Platelets for Part 3
Description: Blood samples were collected for the assessment of hematology parameters namely blood basophils, blood eosinophils, blood leukocytes, blood lymphocytes, blood monocytes, blood neutrophils and blood platelets for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
10^9 cells/liter
  Basophils, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Basophils, Period 1, Day 3 (48 hour), n=10,0,0,2 | 0.004 (0.0158) |  |  | 0.000 (0.0141)
  Basophils, Period 2, Day 3 (48 hour), n=0,10,0,2,: number analyzed (Participants) | 0 | 10 | 0 | 2
  Basophils, Period 2, Day 3 (48 hour), n=0,10,0,2, |  | 0.009 (0.0120) |  | -0.010 (0.0141)
  Basophils, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Basophils, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | 0.009 (0.0162) | 0.005 (0.0071)
  Basophils, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Basophils, Follow-up, n=0,0,9,2 |  |  | 0.008 (0.0186) | 0.015 (0.0071)
  Eosinophils, Period 1, Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Eosinophils, Period 1, Day 3 (48 hour),n=10,0,0,2 | 0.053 (0.0254) |  |  | 0.060 (0.0707)
  Eosinophils, Period 2,Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Eosinophils, Period 2,Day 3 (48 hour), n=0,10,0,2 |  | 0.068 (0.0421) |  | 0.055 (0.0778)
  Eosinophils, Period 3,Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Eosinophils, Period 3,Day 3 (48 hour), n=0,0,9,2 |  |  | 0.053 (0.0487) | 0.040 (0.0990)
  Eosinophils, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Eosinophils, Follow-up, n=0,0,9,2 |  |  | 0.022 (0.0192) | 0.045 (0.1061)
  Leukocytes, Period 1, Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Leukocytes, Period 1, Day 3 (48 hour),n=10,0,0,2 | 0.581 (0.6524) |  |  | -1.000 (0.8202)
  Leukocytes, Period 2, Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Leukocytes, Period 2, Day 3 (48 hour),n=0,10,0,2 |  | 0.730 (0.8427) |  | -1.415 (1.0819)
  Leukocytes, Period 3, Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Leukocytes, Period 3, Day 3 (48 hour),n=0,0,9,2 |  |  | 0.966 (0.7001) | -1.670 (0.9475)
  Leukocytes, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Leukocytes, Follow-up, n=0,0,9,2 |  |  | 0.132 (0.8490) | -1.630 (0.2121)
  Lymphocytes, Period 1,Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Lymphocytes, Period 1,Day 3 (48 hour),n=10,0,0,2 | 0.209 (0.2885) |  |  | 0.060 (0.2263)
  Lymphocytes, Period 2,Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Lymphocytes, Period 2,Day 3 (48 hour),n=0,10,0,2 |  | 0.144 (0.3405) |  | -0.035 (0.2192)
  Lymphocytes, Period 3,Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Lymphocytes, Period 3,Day 3 (48 hour),n=0,0,9,2 |  |  | -0.009 (0.3207) | -0.100 (0.2404)
  Lymphocytes, Follow-up, n=0,0, 9, 2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Lymphocytes, Follow-up, n=0,0, 9, 2 |  |  | -0.089 (0.1928) | -0.050 (0.0283)
  Monocytes, Period 1, Day 3 (48 hour),n=10,0,0,2,: number analyzed (Participants) | 10 | 0 | 0 | 2
  Monocytes, Period 1, Day 3 (48 hour),n=10,0,0,2, | 0.022 (0.0598) |  |  | -0.025 (0.0354)
  Monocytes, Period 2, Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Monocytes, Period 2, Day 3 (48 hour),n=0,10,0,2 |  | 0.010 (0.0615) |  | -0.080 (0.0424)
  Monocytes, Period 3, Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Monocytes, Period 3, Day 3 (48 hour),n=0,0,9,2 |  |  | 0.042 (0.0427) | -0.110 (0.0000)
  Monocytes, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Monocytes, Follow-up, n=0,0,9,2 |  |  | -0.002 (0.0452) | -0.100 (0.0424)
  Neutrophils, Period 1,Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Neutrophils, Period 1,Day 3 (48 hour),n=10,0,0,2 | 0.292 (0.8198) |  |  | -1.100 (1.1597)
  Neutrophils, Period 2,Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Neutrophils, Period 2,Day 3 (48 hour),n=0,10,0,2 |  | 0.489 (0.7302) |  | -1.350 (0.8910)
  Neutrophils, Period 3,Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Neutrophils, Period 3,Day 3 (48 hour),n=0,0,9,2 |  |  | 0.850 (0.8456) | -1.505 (0.7990)
  Neutrophils, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Neutrophils, Follow-up, n=0,0,9,2 |  |  | 0.184 (0.8251) | -1.545 (0.3606)
  Platelets, Period 1, Day 3 (48 hour),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Platelets, Period 1, Day 3 (48 hour),n=10,0,0,2 | -4.7 (13.19) |  |  | -10.5 (10.61)
  Platelets, Period 2, Day 3 (48 hour),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Platelets, Period 2, Day 3 (48 hour),n=0,10,0,2 |  | -22.2 (41.82) |  | -5.0 (5.66)
  Platelets, Period 3, Day 3 (48 hour),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Platelets, Period 3, Day 3 (48 hour),n=0,0,9,2 |  |  | -6.0 (19.80) | -15.0 (8.49)
  Platelets, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Platelets, Follow-up, n=0,0,9,2 |  |  | 2.4 (21.93) | 4.0 (8.49)

102. Secondary Outcome: Change From Baseline in Hematology Parameters Blood Ery. MCHC and Blood Hemoglobin for Part 3
Description: Blood samples were collected for the assessment of hematology parameters namely blood Ery. MCHC and blood hemoglobin for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
grams/liter
  Ery. MCHC, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Ery. MCHC, Period 1, Day 3 (48 hour), n=10,0,0,2 | -2.9 (5.67) |  |  | -2.0 (9.90)
  Ery. MCHC, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Ery. MCHC, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | -3.2 (3.49) |  | -1.5 (4.95)
  Ery. MCHC, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery. MCHC, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | -5.3 (5.22) | -6.5 (2.12)
  Ery. MCHC, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery. MCHC, Follow-up, n=0,0,9,2 |  |  | -1.2 (4.94) | 0.0 (0.00)
  Hemoglobin, Period 1,Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Hemoglobin, Period 1,Day 3 (48 hour), n=10,0,0,2 | -1.4 (6.70) |  |  | -7.5 (0.71)
  Hemoglobin, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Hemoglobin, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | -3.4 (9.35) |  | -11.5 (0.71)
  Hemoglobin, Period 3,Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Hemoglobin, Period 3,Day 3 (48 hour), n=0,0,9,2 |  |  | -2.1 (6.47) | -10.5 (0.71)
  Hemoglobin, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Hemoglobin, Follow-up, n=0,0,9,2 |  |  | -6.0 (7.62) | -6.5 (7.78)

103. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. MCH for Part 3
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCH for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
picograms
  Ery.MCH, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Ery.MCH, Period 1, Day 3 (48 hour), n=10,0,0,2 | 0.08 (0.397) |  |  | 0.25 (0.071)
  Ery.MCH, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Ery.MCH, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | 0.08 (0.270) |  | 0.15 (0.212)
  Ery.MCH, Period 3 Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery.MCH, Period 3 Day 3 (48 hour), n=0,0,9,2 |  |  | -0.12 (0.380) | 0.00 (0.283)
  Ery. MCH, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery. MCH, Follow-up, n=0,0,9,2 |  |  | 0.31 (0.483) | 0.00 (0.424)

104. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. Mean Corpuscular Volume (MCV) for Part 3
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. MCV for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
femtoliters
  Ery. MCV, Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Ery. MCV, Period 1, Day 3 (48 hour), n=10,0,0,2 | 1.10 (1.152) |  |  | 1.30 (2.970)
  Ery. MCV, Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Ery. MCV, Period 2, Day 3 (48 hour), n=0,10,0,2 |  | 1.14 (0.857) |  | 0.70 (2.121)
  Ery. MCV, Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery. MCV, Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | 1.16 (1.167) | 1.80 (0.000)
  Ery. MCV, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery. MCV, Follow-up, n=0,0,9,2 |  |  | 1.31 (1.430) | 0.00 (1.131)

105. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Ery. for Part 3
Description: Blood samples were collected for the assessment of hematology parameter namely blood Ery. for Part 1a. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
10^12 cells/liter
  Ery., Period 1, Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Ery., Period 1, Day 3 (48 hour), n=10,0,0,2 | -0.065 (0.2576) |  |  | -0.275 (0.0354)
  Ery.,Period 2, Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Ery.,Period 2, Day 3 (48 hour), n=0,10,0,2 |  | -0.138 (0.3381) |  | -0.390 (0.0566)
  Ery., Period 3, Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery., Period 3, Day 3 (48 hour), n=0,0,9,2 |  |  | -0.060 (0.2536) | -0.340 (0.0566)
  Ery., Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Ery., Follow-up, n=0,0,9,2 |  |  | -0.253 (0.3347) | -0.210 (0.3111)

106. Secondary Outcome: Change From Baseline in Hematology Parameter Blood Hematocrit for Part 3
Description: Blood samples were collected for the assessment of hematology parameter namely blood hematocrit for Part 3. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
Percentage of red blood cells in blood
  Hematocrit, Period 1,Day 3 (48 hour), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Hematocrit, Period 1,Day 3 (48 hour), n=10,0,0,2 | -0.02 (2.170) |  |  | -2 (0.990)
  Hematocrit, Period 2,Day 3 (48 hour), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Hematocrit, Period 2,Day 3 (48 hour), n=0,10,0,2 |  | -0.65 (2.991) |  | -3.3 (0.424)
  Hematocrit, Period 3,Day 3 (48 hour), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Hematocrit, Period 3,Day 3 (48 hour), n=0,0,9,2 |  |  | 0.02 (2.299) | -2.35 (0.495)
  Hematocrit, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Hematocrit, Follow-up, n=0,0,9,2 |  |  | -1.67 (2.545) | -1.95 (2.333)

107. Secondary Outcome: Change From Baseline in Vital Sign Parameters SBP and DBP for Part 3
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included SBP, DBP. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety population
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
millimeters of mercury
  SBP, Period 1, Day 1 (2 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  SBP, Period 1, Day 1 (2 hours), n=10,0,0,2 | 4.6 (10.94) |  |  | 6.0 (7.07)
  SBP, Period 1, Day 2 (24 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  SBP, Period 1, Day 2 (24 hours), n=10,0,0,2 | -4.3 (11.13) |  |  | 0.5 (3.54)
  SBP, Period 1, Day 3 (48 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  SBP, Period 1, Day 3 (48 hours), n=10,0,0,2 | -4.8 (8.63) |  |  | -1.5 (0.71)
  SBP, Period 2, Day 1 (2 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  SBP, Period 2, Day 1 (2 hours), n=0,10,0,2 |  | 3.5 (11.18) |  | 10.5 (6.36)
  SBP, Period 2, Day 2 (24 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  SBP, Period 2, Day 2 (24 hours), n=0,10,0,2 |  | -2.0 (9.71) |  | 6.0 (7.07)
  SBP, Period 2, Day 3 (48 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  SBP, Period 2, Day 3 (48 hours), n=0,10,0,2 |  | 1.2 (9.37) |  | -3.5 (4.95)
  SBP, Period 3, Day 1 (2 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  SBP, Period 3, Day 1 (2 hours), n=0,0,9,2 |  |  | 7.4 (12.89) | -1.0 (1.41)
  SBP, Period 3, Day 2 (24 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  SBP, Period 3, Day 2 (24 hours), n=0,0,9,2 |  |  | 4.1 (8.19) | -0.5 (2.12)
  SBP, Period 3, Day 3 (48 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  SBP, Period 3, Day 3 (48 hours), n=0,0,9,2 |  |  | -0.7 (10.65) | 0.0 (12.73)
  SBP, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  SBP, Follow-up, n=0,0,9,2 |  |  | 5.1 (7.42) | -4.5 (3.54)
  DBP, Period 1, Day 1 (2 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  DBP, Period 1, Day 1 (2 hours), n=10,0,0,2 | 3.4 (9.63) |  |  | 5.0 (8.49)
  DBP, Period 1, Day 2 (24 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  DBP, Period 1, Day 2 (24 hours), n=10,0,0,2 | -4.4 (7.56) |  |  | 0.0 (7.07)
  DBP, Period 1, Day 3 (48 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  DBP, Period 1, Day 3 (48 hours), n=10,0,0,2 | -3.7 (7.73) |  |  | 2.0 (2.83)
  DBP, Period 2, Day 1 (2 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  DBP, Period 2, Day 1 (2 hours), n=0,10,0,2 |  | -3.4 (7.73) |  | -4.5 (0.71)
  DBP, Period 2, Day 2 (24 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  DBP, Period 2, Day 2 (24 hours), n=0,10,0,2 |  | -2.6 (8.97) |  | -4.0 (0.00)
  DBP, Period 2, Day 3 (48 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  DBP, Period 2, Day 3 (48 hours), n=0,10,0,2 |  | 0.7 (8.81) |  | -4.5 (0.71)
  DBP, Period 3, Day 1 (2 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  DBP, Period 3, Day 1 (2 hours), n=0,0,9,2 |  |  | -2.8 (13.58) | 4.0 (9.90)
  DBP, Period 3, Day 2 (24 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  DBP, Period 3, Day 2 (24 hours), n=0,0,9,2 |  |  | -3.2 (3.96) | 4.0 (0.00)
  DBP, Period 3, Day 3 (48 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  DBP, Period 3, Day 3 (48 hours), n=0,0,9,2 |  |  | -1.3 (9.34) | 3.0 (5.66)
  DBP, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  DBP, Follow-up, n=0,0,9,2 |  |  | 2.2 (9.80) | 2.5 (3.54)

108. Secondary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part 3
Description: Single vital signs were measured in semi-supine position after 5 minutes rest and included heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
beats/minute
  Heart rate, Period 1, Day 1 (2 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Heart rate, Period 1, Day 1 (2 hours), n=10,0,0,2 | 1.6 (8.88) |  |  | 1.0 (15.56)
  Heart rate, Period 2, Day 2 (24 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Heart rate, Period 2, Day 2 (24 hours), n=10,0,0,2 | 0.1 (7.37) |  |  | -4.5 (16.26)
  Heart rate, Period 1, Day 3 (48 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  Heart rate, Period 1, Day 3 (48 hours), n=10,0,0,2 | -3.2 (8.27) |  |  | -4.0 (15.56)
  Heart rate, Period 2, Day 1 (2 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Heart rate, Period 2, Day 1 (2 hours), n=0,10,0,2 |  | 4.9 (6.47) |  | 5.0 (8.49)
  Heart rate, Period 2, Day 2 (24 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Heart rate, Period 2, Day 2 (24 hours), n=0,10,0,2 |  | 0.9 (4.89) |  | 2.0 (7.07)
  Heart rate, Period 2, Day 3 (48 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  Heart rate, Period 2, Day 3 (48 hours), n=0,10,0,2 |  | 3.0 (4.35) |  | -2.5 (0.71)
  Heart rate, Period 3, Day 1 (2 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Heart rate, Period 3, Day 1 (2 hours), n=0,0,9,2 |  |  | 4.6 (7.65) | 7.0 (11.31)
  Heart rate, Period 3, Day 2 (24 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Heart rate, Period 3, Day 2 (24 hours), n=0,0,9,2 |  |  | 1.1 (6.27) | 0.5 (3.54)
  Heart rate, Period 3, Day 3 (48 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Heart rate, Period 3, Day 3 (48 hours), n=0,0,9,2 |  |  | 3.2 (9.92) | 6.5 (12.02)
  Heart rate, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  Heart rate, Follow-up, n=0,0,9,2 |  |  | -4.2 (8.83) | 0.5 (0.71)

109. Secondary Outcome: Change From Baseline in ECG Parameter Heart Rate for Part 3
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that automatically calculated the heart rate. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
beats/minute
  ECG Heart rate,Period1,Day 1 (2 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  ECG Heart rate,Period1,Day 1 (2 hours),n=10,0,0,2 | 8.0 (7.15) |  |  | 5.0 (8.49)
  ECG Heart rate,Period1,Day 2 (24 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  ECG Heart rate,Period1,Day 2 (24 hours),n=10,0,0,2 | -0.3 (4.11) |  |  | -4.0 (4.24)
  ECG Heart rate,Period1,Day 3 (48 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  ECG Heart rate,Period1,Day 3 (48 hours),n=10,0,0,2 | 4.8 (6.75) |  |  | 0.0 (9.90)
  ECG Heart rate,Period2,Day 1 (2 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  ECG Heart rate,Period2,Day 1 (2 hours),n=0,10,0,2 |  | 6.4 (8.88) |  | 10.0 (7.07)
  ECG Heart rate,Period2,Day 2 (24 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  ECG Heart rate,Period2,Day 2 (24 hours),n=0,10,0,2 |  | -0.2 (8.78) |  | 8.0 (8.49)
  ECG Heart rate,Period2,Day 3 (48 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  ECG Heart rate,Period2,Day 3 (48 hours),n=0,10,0,2 |  | -0.5 (10.32) |  | 3.0 (5.66)
  ECG Heart rate,Period3,Day 1 (2 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  ECG Heart rate,Period3,Day 1 (2 hours),n=0,0,9,2 |  |  | 8.0 (7.04) | 5.5 (6.36)
  ECG Heart rate,Period3,Day 2 (24 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  ECG Heart rate,Period3,Day 2 (24 hours),n=0,0,9,2 |  |  | 4.6 (13.61) | 12.0 (15.56)
  ECG Heart rate,Period3,Day 3 (48 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  ECG Heart rate,Period3,Day 3 (48 hours),n=0,0,9,2 |  |  | 1.4 (5.98) | 5.0 (9.90)
  ECG Heart rate, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  ECG Heart rate, Follow-up, n=0,0,9,2 |  |  | -3.8 (6.72) | -1.0 (0.00)

110. Secondary Outcome: Change From Baseline in ECG Parameters PR Interval, QRS Duration, QT Interval, QTcB and QTcF for Part 3
Description: A 12 lead ECG was measured in semi-supine position after 5 minutes rest using an ECG machine that measured PR interval, QRS duration, QT interval, QTcB and QTcF for Part 3. Baseline was defined as assessments performed on Day 1 (pre-dose). Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Time Frame: Baseline and up to 14 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
milliseconds
  PR interval, Period1,Day 1 (2 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  PR interval, Period1,Day 1 (2 hours),n=10,0,0,2 | -3.3 (12.58) |  |  | -1.0 (5.66)
  PR interval, Period1,Day 2 (24 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  PR interval, Period1,Day 2 (24 hours),n=10,0,0,2 | -1.9 (7.82) |  |  | -1.0 (5.66)
  PR interval,Period1,Day 3 (48 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  PR interval,Period1,Day 3 (48 hours), n=10,0,0,2 | -3.7 (9.08) |  |  | 0.0 (4.24)
  PR interval,Period 2,Day 1 (2 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  PR interval,Period 2,Day 1 (2 hours),n=0,10,0,2 |  | -7.5 (12.70) |  | -8.5 (0.71)
  PR interval,Period 2, Day 2 (24 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  PR interval,Period 2, Day 2 (24 hours),n=0,10,0,2 |  | -2.2 (9.02) |  | 1.0 (4.24)
  PR interval, Period2, Day 3 (48 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  PR interval, Period2, Day 3 (48 hours),n=0,10,0,2 |  | -3.5 (13.92) |  | 3.0 (1.41)
  PR interval,Period 3,Day 1 (2 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  PR interval,Period 3,Day 1 (2 hours),n=0,0,9,2 |  |  | -0.1 (6.77) | -4.0 (14.14)
  PR interval,Period 3,Day 2 (24 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  PR interval,Period 3,Day 2 (24 hours),n=0,0,9,2 |  |  | 4.8 (13.94) | 0.5 (7.78)
  PR interval,Period 3,Day 3 (48 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  PR interval,Period 3,Day 3 (48 hours), n=0,0,9,2 |  |  | 0.3 (16.18) | 4.0 (16.97)
  PR interval, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  PR interval, Follow-up, n=0,0,9,2 |  |  | 6.1 (11.95) | -6.0 (24.04)
  QRS duration,Period 1,Day 1 (2 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QRS duration,Period 1,Day 1 (2 hours),n=10,0,0,2 | 2.0 (10.73) |  |  | 3.5 (9.19)
  QRS duration,Period 1,Day 2 (24 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QRS duration,Period 1,Day 2 (24 hours),n=10,0,0,2 | 4.3 (8.63) |  |  | -3.0 (7.07)
  QRS duration,Period 1,Day 3 (48 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QRS duration,Period 1,Day 3 (48 hours),n=10,0,0,2 | 0.5 (10.50) |  |  | 2.0 (4.24)
  QRS duration,Period 2,Day 1 (2 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QRS duration,Period 2,Day 1 (2 hours),n=0,10,0,2 |  | 1.8 (4.71) |  | 2.0 (7.07)
  QRS duration,Period 2, Day 2 (24 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QRS duration,Period 2, Day 2 (24 hours),n=0,10,0,2 |  | 0.4 (7.07) |  | -2.5 (19.09)
  QRS duration,Period 2, Day 3 (48 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QRS duration,Period 2, Day 3 (48 hours),n=0,10,0,2 |  | -1.1 (6.40) |  | 1.5 (3.54)
  QRS duration,Period 3,Day 1(2 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QRS duration,Period 3,Day 1(2 hours),n=0,0,9,2 |  |  | 2.9 (4.65) | 1.5 (4.95)
  QRS duration,Period 3,Day 2(24 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QRS duration,Period 3,Day 2(24 hours),n=0,0,9,2 |  |  | -2.6 (4.39) | 8.0 (8.49)
  QRS duration,Period3, Day 3(48 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QRS duration,Period3, Day 3(48 hours),n=0,0,9,2 |  |  | -1.1 (8.74) | 3.5 (14.85)
  QRS duration, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QRS duration, Follow-up, n=0,0,9,2 |  |  | -0.7 (6.52) | 4.5 (7.78)
  QT interval,Period 1, Day 1(2 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QT interval,Period 1, Day 1(2 hours),n=10,0,0,2 | -9.2 (19.47) |  |  | -15.0 (19.80)
  QT interval,Period 1,Day 2(24 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QT interval,Period 1,Day 2(24 hours),n=10,0,0,2 | 7.9 (19.45) |  |  | -6.0 (24.04)
  QT interval,Period 1, Day 3(48 hours),n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QT interval,Period 1, Day 3(48 hours),n=10,0,0,2 | 0.4 (22.89) |  |  | -0.5 (12.02)
  QT interval,Period 2, Day 1 (2 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QT interval,Period 2, Day 1 (2 hours),n=0,10,0,2 |  | -4.0 (22.45) |  | -14.5 (23.33)
  QT interval,Period 2, Day 2 (24 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QT interval,Period 2, Day 2 (24 hours),n=0,10,0,2 |  | 3.7 (15.93) |  | -12.5 (31.82)
  QT interval,Period 2, Day 3 (48 hours),n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QT interval,Period 2, Day 3 (48 hours),n=0,10,0,2 |  | 0.0 (26.86) |  | -3.0 (2.83)
  QT interval,Period 3, Day 1 (2 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QT interval,Period 3, Day 1 (2 hours),n=0,0,9,2 |  |  | -7.9 (11.61) | -12.5 (31.82)
  QT interval,Period 3, Day 2 (24 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QT interval,Period 3, Day 2 (24 hours),n=0,0,9,2 |  |  | -6.2 (24.03) | -15.0 (28.28)
  QT interval,Period 3, Day 3 (48 hours),n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QT interval,Period 3, Day 3 (48 hours),n=0,0,9,2 |  |  | -3.0 (15.28) | -15.0 (36.77)
  QT interval, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QT interval, Follow-up, n=0,0,9,2 |  |  | 11.4 (17.84) | 8.5 (6.36)
  QTcB ,Period 1, Day 1 (2 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QTcB ,Period 1, Day 1 (2 hours), n=10,0,0,2 | 16.4 (25.48) |  |  | -1.0 (2.83)
  QTcB, Period 1, Day 2 (24 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QTcB, Period 1, Day 2 (24 hours), n=10,0,0,2 | 8.6 (16.10) |  |  | -19.5 (9.19)
  QTcB, Period 1, Day 3 (48 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QTcB, Period 1, Day 3 (48 hours), n=10,0,0,2 | 15.7 (14.70) |  |  | -1.0 (19.80)
  QTcB, Period 2, Day 1 (2 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QTcB, Period 2, Day 1 (2 hours), n=0,10,0,2 |  | 15.1 (20.18) |  | 15.0 (8.49)
  QTcB, Period 2, Day 2 (24 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QTcB, Period 2, Day 2 (24 hours), n=0,10,0,2 |  | 5.1 (13.98) |  | 9.5 (12.02)
  QTcB, Period 2, Day 3 (48 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QTcB, Period 2, Day 3 (48 hours), n=0,10,0,2 |  | 1.8 (12.99) |  | 5.5 (13.44)
  QTcB, Period 3, Day 1 (2 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcB, Period 3, Day 1 (2 hours), n=0,0,9,2 |  |  | 14.9 (21.83) | 4.0 (14.14)
  QTcB, Period 3, Day 2 (24 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcB, Period 3, Day 2 (24 hours), n=0,0,9,2 |  |  | 5.8 (11.14) | 18.5 (12.02)
  QTcB, Period 3, Day 3 (48 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcB, Period 3, Day 3 (48 hours), n=0,0,9,2 |  |  | 2.1 (10.02) | -3.0 (8.49)
  QTcB, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcB, Follow-up, n=0,0,9,2 |  |  | 1.9 (14.88) | 6.5 (6.36)
  QTcF, Period 1, Day 1 (2 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QTcF, Period 1, Day 1 (2 hours), n=10,0,0,2 | 7.7 (20.94) |  |  | -6.0 (5.66)
  QTcF, Period 1, Day 2 (24 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QTcF, Period 1, Day 2 (24 hours), n=10,0,0,2 | 8.3 (16.09) |  |  | -15.0 (14.14)
  QTcF, Period 1, Day 3 (48 hours), n=10,0,0,2: number analyzed (Participants) | 10 | 0 | 0 | 2
  QTcF, Period 1, Day 3 (48 hours), n=10,0,0,2 | 10.5 (14.75) |  |  | -1.0 (8.49)
  QTcF, Period 2, Day 1 (2 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QTcF, Period 2, Day 1 (2 hours), n=0,10,0,2 |  | 8.4 (17.65) |  | 5.0 (14.14)
  QTcF, Period 2, Day 2 (24 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QTcF, Period 2, Day 2 (24 hours), n=0,10,0,2 |  | 4.5 (7.09) |  | 2.5 (19.09)
  QTcF, Period 2, Day 3 (48 hours), n=0,10,0,2: number analyzed (Participants) | 0 | 10 | 0 | 2
  QTcF, Period 2, Day 3 (48 hours), n=0,10,0,2 |  | 1.2 (10.25) |  | 2.5 (7.78)
  QTcF, Period 3, Day 1 (2 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcF, Period 3, Day 1 (2 hours), n=0,0,9,2 |  |  | 6.8 (16.15) | -1.5 (20.51)
  QTcF, Period 3, Day 2 (24 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcF, Period 3, Day 2 (24 hours), n=0,0,9,2 |  |  | 1.2 (4.99) | 7.0 (2.83)
  QTcF, Period 3, Day 3 (48 hours), n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcF, Period 3, Day 3 (48 hours), n=0,0,9,2 |  |  | 0.2 (9.18) | -7.0 (18.38)
  QTcF, Follow-up, n=0,0,9,2: number analyzed (Participants) | 0 | 0 | 9 | 2
  QTcF, Follow-up, n=0,0,9,2 |  |  | 5.2 (13.55) | 7.0 (7.07)

111. Secondary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Analysis Part 3
Description: Urinalysis parameters assessed were urine ketones, urine glucose, urine occult blood, urine pH, urine specific gravity and urine protein. In this dipstick test, the level of ketones, glucose, occult blood, pH, specific gravity and protein in urine samples was recorded as negative trace, 1+, 3+, 5+, 6+, 7+ and 8+ (the plus sign increases with a higher level of ketones, occult blood, pH or specific gravity in the urine: 1+=slightly positive, 3+ to 5+=positive, 6+ and above=high positive). Urine samples were collected for the measurement of urinalysis parameters by dipstick method up-to follow-up (5 to 7 days post last dose) in Part 3. Only categories with significant values have been presented.
Time Frame: Up to 14 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
Number analyzed (Participants) | 10 | 10 | 9 | 2
Participants
  Urine Ketones, Follow-up, 1+ | 0 | 0 | 1 | 0
  Urine Occult blood,Trace,Period 1, Day 3 (48hours) | 2 | 0 | 0 | 0
  Urine Occult blood,Period 1,Day 3 (48hours), 1+ | 0 | 0 | 0 | 1
  Urine Occult blood,Period 1,Day 3 (48hours), 3+ | 1 | 0 | 0 | 0
  Urine Occult blood,Trace,Period 2,Day 3 (48hours) | 0 | 1 | 0 | 0
  Urine Occult blood,Period 2,Day 3 (48hours), 1+ | 0 | 1 | 0 | 0
  Urine Occult blood,Trace,Period 3,Day 3 (48hours) | 0 | 0 | 2 | 0
  Urine Occult blood,Period 3,Day 3 (48hours), 1+ | 0 | 0 | 1 | 0
  Urine Occult blood, Follow-up, 4+ | 0 | 0 | 1 | 0
  Urine pH, Period 1 Day 3 (48 hours), 5+ | 0 | 0 | 0 | 1
  Urine pH, Period 1, Day 3 (48 hours), 6+ | 4 | 0 | 0 | 1
  Urine pH, Period 1, Day 3 (48 hours), 7+ | 5 | 0 | 0 | 1
  Urine pH, Period 1, Day 3 (48 hours), 8+ | 1 | 0 | 0 | 0
  Urine pH, Period 2, Day 3 (48 hours), 5+ | 0 | 6 | 0 | 2
  Urine pH, Period 2, Day 3 (48 hours), 6+ | 0 | 2 | 0 | 0
  Urine pH, Period 2, Day 3 (48 hours), 7+ | 0 | 2 | 0 | 0
  Urine pH, Period 3, Day 3 (48 hours), 5+ | 0 | 0 | 3 | 0
  Urine pH, Period 3, Day 3 (48 hours), 6+ | 0 | 0 | 5 | 2
  Urine pH, Period 3, Day 3 (48 hours), 7+ | 0 | 0 | 1 | 0
  Urine pH, Follow-up, 5+ | 0 | 0 | 3 | 1
  Urine pH, Follow-up, 6+ | 0 | 0 | 2 | 1
  Urine pH, Follow-up, 7+ | 0 | 0 | 4 | 0
  Urine Specific gravity, Period1,Day 3(48 hours),1+ | 10 | 0 | 0 | 2
  Urine Specific gravity, Period2,Day 3(48 hours),1+ | 0 | 10 | 0 | 2
  Urine Specific gravity,Period 3,Day 3(48 hours),1+ | 0 | 0 | 9 | 2
  Urine Specific gravity, Follow-up, 1+ | 0 | 0 | 9 | 2

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from Day 1 until follow-up (Up to 14 days in Part 1a, 11 days in Part 1b and 2 and 14 days in Part 3).
Description: Safety population was used to assess non-serious AEs and SAEs.
Groups:
- Gepotidacin 1500 mg - R Capsules: Participants received gepotidacin 1500 mg (3 x 500) mg - R capsules orally in one of the 3 treatment periods for 3 days in Part 1a.
- Gepotidacin 1500 mg RC Tablets: Participants received gepotidacin 1500 mg (2 x 750) RC tablets orally in one of the 3 treatment periods for 3 days in Part 1a.
- Gepotidacin 1500 mg HSWG Tablets: Participants received gepotidacin 1500 mg (2 x 750) HSWG tablets orally in one of the three treatment periods in Part 1a.
- Gepotidacin RC 1500 mg Tablets; Gepotidacin RC 3000 mg Tablets: Participants received a single dose gepotidacin 3000 mg (4 x 750 mg) RC tablets orally in Part 2 Period 2.
- Gepotidacin RC 1500 mg Fed; Gepotidacin RC 2250 mg Fed: Participants received gepotidacin 1500 mg (2 x 750) RC tablets in the fed state orally in one of the 3 treatment periods for 3 days in Part 3.
- Gepotidacin RC 3000 mg Fed: Participants received gepotidacin 3000 mg (4 x 750) RC tablets in the fed state in one of the 3 treatment periods in Part 3.
Arm/Group | Gepotidacin 1500 mg - R Capsules | Gepotidacin 1500 mg RC Tablets | Gepotidacin 1500 mg HSWG Tablets | Gepotidacin RC 1500 mg Tablets | Gepotidacin RC 3000 mg Tablets | Gepotidacin RC 1500 mg Fed | Gepotidacin RC 2250 mg Fed | Gepotidacin RC 3000 mg Fed | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/10 | 0/10 | 0/10 | 0/10 | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/10 | 0/10 | 0/10 | 0/10 | 0/9 | 0/2
Other Adverse Events (participants affected / at risk) | 8/26 | 5/26 | 9/26 | 6/10 | 9/10 | 0/10 | 1/10 | 6/9 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gepotidacin 1500 mg - R Capsules (N=26) | Gepotidacin 1500 mg RC Tablets (N=26) | Gepotidacin 1500 mg HSWG Tablets (N=26) | Gepotidacin RC 1500 mg Tablets (N=10) | Gepotidacin RC 3000 mg Tablets (N=10) | Gepotidacin RC 1500 mg Fed (N=10) | Gepotidacin RC 2250 mg Fed (N=10) | Gepotidacin RC 3000 mg Fed (N=9) | Placebo (N=2)
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 6 | 5 | 9 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 6 | 0 | 0 | 4 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 2 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02853435/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT02853435/SAP_001.pdf